

# UNIVERSITY OF VERMONT CENTER ON TOBACCO REGULATORY SCIENCE

# PROJECT 2, STUDY 3

### LOW NICOTINE CONTENT CIGARETTES IN VULNERABLE POPULATIONS: OPIOID USE DISORDER

STUDY PROTOCOL

Version 34: 9 December 2022

# CHRMS (Medical) #19-0130 Approved: 1/23/2023



| Table of Contents | |
|---|---|
| 1. Objective6 | 3 |
| 2. Significance | 7 |
| 2.1 Opioid Use Disorder (OUD) and smoking | 7 |
| 2.2 Reducing the addiction potential of tobacco products. | 8 |
| 2.3 Relevance of the project to the integrative theme and goals of the TCORS | 8 |
| 2.4 Relevance to the scientific domains and priorities of the FDA CTP. | 8 |
| 2.5 How study outcomes will improve scientific knowledge related to the manufacture, distribution and marketing of tobacco products | |
| 3. Rationale | 9 |
| 3.1 Effects of nicotine reduction in smokers with OUD. | 9 |
| 3.2 Increasing appeal of alternative non-combusted nicotine sources | 0 |
| 3.3 E-cig use11 | 1 |
| 3.4 E-cig effects on smoking11 | 1 |
| 3.5 Importance of e-cig flavors1 | 1 |
| 3.6 Products to be tested | 2 |
| 3.7 Summary | 2 |
| 4. Project Study Methods12 | 2 |
| 5. Study Screening Procedures | 3 |
| 5.1 Participants1 | 3 |
| 5.2 Recruitment13 | 3 |
| 5.3 Informed Consent Process15 | 5 |
| 5.4 Screening Measures15 | 5 |
| 5.5 Suicidality/Mental Health Monitoring17 | 7 |
| 5.6 Inclusion/Exclusion Criteria17 | 7 |
| 5.7 Eligibility Determination20 | J |
| 6 Study Baseline Procedures | ሰ |

# CHRMS (Medical) #19-0130 Approved: 1/23/2023



| 6.1 Visit scheduling requirements for baseline period | 21 |
|---|---|
| 6.2 Measures/Assessments | 22 |
| 6.3 E-Cigarette Training session | 24 |
| 6.4 Interactive Voice Response | 24 |
| 7. Study Experimental Procedures. | 25 |
| 7.1 Experimental Period | 25 |
| 7.2 Experimental Visits Weeks 1, 3, 5, 7, 9, 11, 13 and 15 Procedures | 26 |
| 7.2.A Measures/ Assessments | 26 |
| 7.3 Experimental Visits Weeks 2, 4, 6, 8, 10, 12, 14 and 16 Procedures | 26 |
| 7.3.A Measures/Assessments | 26 |
| 7.4 Interactive Voice Response System. | 27 |
| 7.5 Variable Incentive Program. | 28 |
| 7.6 Product and Procedures Compliance Review Sessions. | 29 |
| 7.7 Quit Attempts During the Study Protocol | 29 |
| 7.7.A If a Participant is Currently Abstaining from Smoking with the Intention Quit. | |
| 7.7.B If a Participant is Planning to Quit Smoking, but has not initiated the q attempt | |
| 7.8 Abstinence Assessment Session. | 30 |
| 7.8.A Participants Who Meet Criteria for Abstinence | 30 |
| 7.8.A.1 Measures/Assessments | 30 |
| 7.8.B Participants Who Do Not Meet Criteria for Abstinence | 31 |
| 7.8.B.1 Measures/Assessments | 31 |
| 7.9. Participant Compensation | 31 |
| 7.10 End of Study. | 32 |
| 7.11 30 Day Follow up Phone Call. | 32 |
| 8. Study Randomization | 33 |

# CHRMS (Medical) #19-0130 Approved: 1/23/2023



| 8.1 Randomization Process. | 33 |
|---------------------------------------------------------|----|
| 8.2 Study Product Administration. | 33 |
| 8.3 Guidelines for Reporting Other Nicotine Product Use | 33 |
| 8.4 Study Product Accountability | 34 |
| 9. Study 3 Statistical Methods and Sample Size. | 34 |
| 9.1 Statistical Methods. | 34 |
| 9.2 Sample Size | 35 |
| 10. Potential Risks of Participation | 36 |
| 10.1 Risks of Participation | 36 |
| 10.2 Avoiding Risk to Fetus. | 38 |
| 10.3 Expected benefits of participation | 38 |
| 11. Protection Against Risk | 38 |
| 11.1 Data Collection Protections. | 38 |
| 11.2 Data Storage | 39 |
| 12. Adverse Events. | 39 |
| 13. Withdrawal or Monitoring of Participants. | 40 |
| 14. Data Safety Monitoring Board | 41 |
| 15. Investigational Tobacco Product | 42 |
| 16. Certificate of Confidentiality. | 42 |
| 17. Outcome Variables. | 43 |
| 18. References. | 44 |



#### **Abbreviations**

- 3HC: 3-hydroxycotinine
- BAL: Breath alcohol levels
- BDI: Beck's Depression Inventory
- BMI: Body Mass Index
- BP: Blood pressure
- BPM: Beats per minute
- BRIEF-A: Behavioral Rating Inventory of Executive Function
- CES: Cigarette Evaluation Scale
- CO: Carbon monoxide
- COT: Cotinine
- CPD: Cigarettes per day
- CPT: Cigarette Purchase Task
- CPT: Continuous Performance Task
- DAST: Drug Abuse Screening Test
- DDT: Delay Discounting Task
- D-KEFS: Delis-Kaplan Executive Function System
- EDC: Electronic Data Capture
- EQ-5D: Euro-Qol
- FSPTCA: Family Smoking Prevention and Tobacco Control Act
- FTND: Fagerström Test for Nicotine Dependence
- GAD: Generalized Anxiety Disorder
- HR: Heart rate
- IVR: Interactive Voice Response
- MDD: Major Depressive Disorder
- MINI: Mini International Neuropsychiatric Interview
- MNWS: Minnesota Nicotine Withdrawal Scale
- NMR: Nicotine metabolite ratio
- NNAL: 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol
- NNC: Normal nicotine content
- NNN: N'-nitrosonornicotine
- OASIS: Overall Anxiety Severity and Impairment Scale
- OUD: Opioid Use Disorder
- PANAS: Positive and Negative Affect Schedule
- PHQ: Patient Health Questionnaire
- PSS: Perceived Stress Scale
- QSU: Questionnaire of Smoking Urges
- RNC: Reduced nicotine content
- SST: Stop Signal Task
- TLFB: Timeline Follow Back
- TPQ: Time Perspectives Questionnaire
- VLNC: Very low nicotine content
- WASI-II: Wechsler Abbreviated Scale of Intelligence-II
- WISDM: Wisconsin Index of Smoking Dependence Motives



# **Project 2 Protocol**

#### 1. OBJECTIVE

Prevalence of smoking among individuals with opioid use disorder (OUD) is six-fold that of the general US adult population. The mortality rate of opioid-dependent smokers is four times that of opioid-dependent nonsmokers, and their response to smoking cessation interventions is notoriously poor. A national policy of reducing the nicotine content of cigarettes has the potential to be an effective method of reducing tobacco use prevalence, dependence, and related adverse health outcomes. Controlled trials in the general smoker population have demonstrated that switching smokers to very low nicotine content cigarettes (VLNCCs) results in reductions in cigarettes per day (CPD), dependence and tobacco toxicant exposure, with few adverse consequences. Furthermore, our work during the current funding period indicates that smokers with OUD also respond to reductions in cigarette nicotine content with reductions in cigarette demand and other measures of addiction potential, although to a lesser extent than the other vulnerable smoker populations we have been examining (i.e., economically disadvantaged women, individuals with affective disorders). We believe that the impact of reduced nicotine standards on use of combusted cigarettes in this highly tobacco addicted population will be moderated considerably by other tobacco market conditions including (1) availability of alternative sources of non-combusted nicotine, and (2) whether these alternatives are available under conditions that optimize their appeal. We hypothesize the same for other vulnerable populations as well, but achieving significant reductions in use of combusted cigarettes in smokers with OUD seems especially unlikely in the absence of readily available and appealing alternative sources of non-combusted nicotine.

The goal of the proposed trial is to experimentally model whether increased availability and appeal of an alternative, non-combusted source of nicotine (e-cigarettes) will enhance the effectiveness of a reduced nicotine standard for cigarettes in smokers with OUD. Daily smokers receiving methadone or buprenorphine treatment will be recruited at University of Vermont and Johns Hopkins University and randomized to one of the following conditions: (1) normal nicotine content cigarettes (NNCC) alone, serving as the control condition, (2) VLNCCs alone, (3) VLNCCs + tobacco-flavored nicotinized e-cigarettes (TF e-cigs), or (4) VLNCCs + nicotinized e-cigarette with preferred flavoring (PF e-cigs). Participants will be asked to use only their assigned products for 16 weeks. Outcome measures include total CPD, product demand using behavioral-economic purchase tasks, craving, withdrawal, and biomarkers of tobacco toxicant exposure. In Week 17, participants will abstain from combusted cigarette use and we will assess effects on cigarette craving, withdrawal and demand.

This research will address the following specific aims:

Aim 1 (Primary): To compare the effects of: (1) NNCCs alone, (2) VLNCCs alone, (3) VLNCCs + TF e-cigs and (4) VLNCCs + PF e-cigs on total CPD in smokers with OUD. We hypothesize that at Week 16, total CPD will be reduced in a linear manner, with the largest reduction in the VLNCCs + PF e-cig condition.

Aim 2 (Secondary): To compare the effects of study conditions on measures of cigarette demand, smoke exposure (breath CO) and tobacco carcinogen biomarkers (NNAL, PAHs) in smokers with OUD. We hypothesize that at Week 16, these measures will have decreased in a linear manner, with the largest reduction in the VLNCCs + PF e-cig condition.

Aim 3 (Exploratory): To explore the effects of the four study conditions on cigarette demand,



craving, and withdrawal in smokers with OUD during the abstinence assessment period.

The integrative theme of this TCORS is vulnerable populations. The proposed research is relevant to FDA CTP's scientific domains of Addiction and Behavior by addressing whether reducing the nicotine content of cigarettes reduces cigarette use, dependence, and product appeal, and whether these effects are enhanced by availability of appealing alternative sources of non-combusted nicotine. It addresses the domain of Health Effects by assessing tobacco toxicant exposure and other biomarkers. The proposed study is significant and innovative by modeling the potential moderating effects of e-cigarette availability and appeal on a national reduced-nicotine policy for cigarettes in this understudied population. Finally, it is programmatic as it builds directly upon and extends the work our team accomplished during the Phase 1 funding period

#### 2. SIGNIFICANCE

# 2.1. Opioid Use Disorder (OUD) and smoking

Cigarette smoking is the leading preventable cause of US morbidity and mortality.¹ While smoking has steadily declined in the general population, it remains entrenched among vulnerable populations. Individuals with substance use disorders, mental illness or socioeconomic disadvantage are disproportionately represented among current cigarette smokers and bear a disproportionate burden of smoking attributable disease and premature death.²-⁵ The focus of this proposal is on the vulnerable population of smokers with concurrent substance abuse. Recent data from Wave 1 of the Population Assessment of Tobacco and Health study show that among current adult cigarette smokers, 80.7% report past-year alcohol or drug use.⁶ Current smokers are more than twice as likely as non-smokers to report past-year misuse of painkillers/sedatives and more than four times as likely to be past-year users of other drugs, including heroin. Conversely, individuals with substance use disorders (SUDs) are substantially more likely to die of tobacco-related disorders (e.g., lung and larynx cancers, respiratory disease) than the general population.<sup>7-9</sup> They are also more likely to die of problems related to their tobacco use than other drug use.<sup>10</sup>

As an exemplar of the larger population of smokers with SUDs, we have been focusing on those with concomitant opioid use disorder (OUD). The disproportionate burden of smoking and smoking-related consequences is especially evident in these individuals. Prevalence of smoking among adults with OUD is six-fold that of the general US adult population (84-94% vs. 15%, respectively). Smokers with OUD also have greater severity of nicotine dependence. In recent analyses by our group of data from the National Survey on Drug Use and Health (2006-2014), after accounting for sociodemographic and smoking characteristics, mean Nicotine Dependence Syndrome Scale scores were significantly higher for opioid-dependent smokers vs. smokers not dependent on opioids (p<0.05). Finally, smoking is associated with significant morbidity and mortality in this population, with the mortality rate of opioid-dependent smokers four times that of opioid-dependent nonsmokers. 7,9-10

The majority of OUD patients report knowledge of the adverse health consequences of smoking as well as a desire to quit smoking. 12,16-17,19-23 Despite this, their responses to standard smoking cessation treatments, including standard pharmacotherapies, are notoriously poor, with quit rates one-fourth that of non-substance abusers. 16, 24-29 Taken together, the high smoking prevalence, poor treatment response, and public health costs associated with smoking among opioid-dependent individuals are of significant concern given the scope of the current opioid epidemic, with 5% of Americans - over 16 million people - reporting recent opioid abuse. 30-31



# 2.2. Reducing the addiction potential of tobacco products

One potential way to reduce smoking prevalence is to implement public policy mandating a reduction in cigarette nicotine content below the threshold necessary to establish and sustain nicotine dependence.<sup>32</sup> The 2009 Family Smoking Prevention and Tobacco Control Act gave the FDA the authority to regulate tobacco products to protect public health, including limiting the nicotine content of cigarettes. Nicotine is the constituent in tobacco that drives repeated use, dependence, and eventually the chronic diseases and premature death that result from chronic smoke exposure. Thus, reductions in nicotine content may reduce smoking prevalence and related disease by disrupting initiation of smoking by new users and increasing cessation rates among current smokers.<sup>33-34</sup> This approach could be particularly beneficial to subpopulations of smokers who have less success with currently available cessation treatments, such as people with OUD.<sup>35</sup> Our work during the current funding period, reviewed below, indicates that smokers with OUD respond to reductions in the nicotine content of cigarettes with reductions in cigarette demand and other measures of addiction potential, although to a lesser extent than the other vulnerable smoker populations we have been examining (i.e., economically disadvantaged women, individuals with affective disorders (AD)). We anticipate that a combination of tobacco market conditions will be necessary to produce a maximal effect on combusted smoking in this population. In particular, we hypothesize that (1) making alternative sources of non-combusted nicotine (i.e., electronic cigarettes; e-cigs) available and (2) doing so under conditions that optimize their appeal (i.e., preferred flavoring) may enhance the ability of a national policy to reduce nicotine standards to decrease cigarette smoking, dependence, and related adverse health outcomes among smokers with OUD.

# 2.3. Relevance of the project to the integrative theme and goals of the TCORS

The integrative theme of our UVM TCORS is **vulnerable populations**, and our goals are to model the potential effects of tobacco product standards on product use in vulnerable populations, with the goal of reducing the risks of product use, dependence, and related adverse health outcomes. For the FDA to effectively execute its tobacco regulatory responsibilities, it must have sound scientific evidence on how product standards impact tobacco use in populations with high rates of tobacco dependence. Our goal is to provide the FDA with that evidence. This project is relevant to that goal because it will examine the effects of a reduced-nicotine standard for cigarettes, alone and combined with another FDA-regulated product (e-cigs) on measures of cigarette use, demand, dependence and tobacco toxicant exposure in this vulnerable population.

#### 2.4. Relevance to the scientific domains and priorities of the FDA CTP

The proposed research is highly relevant to the CTP's scientific domains of **Addiction** and **Behavior** because it will address whether reducing the nicotine content of cigarettes reduces cigarette use, dependence, and product appeal, and whether these effects are enhanced by the availability of appealing alternative sources of non-combusted nicotine. It will address the **Health Effects** domain by assessing the effects of these conditions on tobacco toxicant exposure and a respiratory biomarker.

# 2.5. How study outcomes will improve scientific knowledge related to the manufacture, distribution and marketing of tobacco products

Outcomes will directly inform scientific knowledge concerning the manufacture of tobacco products by demonstrating whether a reduction in the maximum nicotine content of cigarettes to  $\leq 0.4$  mg nicotine/g tobacco would reduce smoking in this vulnerable population. The outcomes will also indicate whether continuing to allow the sale of e-cigs in characterizing flavors improves the efficacy of a reduced-nicotine standard for cigarettes on smoking reduction in this population.



#### 3. RATIONALE

#### 3.1. Effects of nicotine reduction in smokers with OUD

There is growing evidence to support the public health benefit of a nicotine reduction policy. Studies in the general smoker population have demonstrated that use of reduced nicotine content cigarettes decreases smoking rates, dependence and toxin exposure levels. 33,36-46 However, these studies were conducted with psychiatrically and socioeconomically stable, healthy smokers. While a national nicotine reduction policy may hold significant potential to reduce smoking prevalence and related adverse health outcomes, it is important to first understand whether vulnerable populations of smokers may respond differently than the general population. 43,47 This includes the possibility that these subgroups respond to reduced nicotine content cigarettes (RNCCs) with compensatory smoking, which could lead to increased carcinogen and other toxin exposure, failure to use RNCCs altogether, or transition to use of other products (e.g., cigars) which would undermine the merit of this regulatory strategy. 48,49

Research conducted by our UVM TCORS provides encouraging evidence that the beneficial effects of very low nicotine content cigarettes (VLNCCs) may extend to populations that are highly vulnerable to tobacco addiction and its associated adverse health consequences. During the current funding period, we have been conducting two multi-site studies examining acute and extended exposure to RNCCs on the addiction potential of smoking. The initial acute exposure study consisted of three parallel, within-subject laboratory studies in economically disadvantaged women of reproductive age (n=56), individuals with OUD (n=60), and individuals with AD (n=53).<sup>50</sup>

Participants sampled NIDA-provided research cigarettes varying in nicotine content (15.8, 2.4, 1.3, 0.4mg/g) under double-blind conditions, with the highest dose representing nicotine content typical of commercial cigarettes. Following brief abstinence, participants completed 14 sessions comparing the relative reinforcing effects of the 6 possible dose pairs in concurrent choice procedures. We also assessed demand for each cigarette dose using the Cigarette Purchase Task (CPT), a behavioral economic task that models hypothetical demand for cigarettes under varying prices. Lastly, we compared cigarettes on smoking topography and subjective effects.

Results were collapsed across populations as similarities outnumbered differences. In concurrent choice testing, participants chose the higher over the lower nicotine content cigarettes across each of the six dose pairs when available at the same low price, providing strong evidence that reducing nicotine content decreases the relative reinforcing effects (i.e., addiction potential) of smoking in a graded dose-dependent manner (Figure 1, upper panel). Importantly in terms of regulatory implications, we also



Figure 1. Concurrent Choice Testing

demonstrated that the robust preference for the high 15.8 mg/g control dose over the 0.4 mg/g dose was reversed in all three populations by incrementing the response effort required to obtain the high dose while keeping the low dose available at the same low response requirement (lower panel). This suggests that product preference is conditional on environmental context. Demand for cigarettes on the CPT task also decreased as an orderly function of nicotine content consistent with the differences in relative reinforcing effects seen in the concurrent choice task. Importantly, there was no evidence of compensatory smoking. This study provided a compelling demonstration that RNCCs reduce the addiction potential of cigarettes in populations highly vulnerable to tobacco addiction. It is worth noting, however, that we observed greater overall



cigarette demand across doses in smokers with OUD vs. the other vulnerable populations examined in this study.

Our second multi-site study is ongoing and on schedule to be completed as planned. The study uses a three parallel-groups design to investigate the effects of 12-week exposure to RNCCs (15.8, 2.4, and 0.4 mg/g). Preliminary results on total cigarettes per day (CPD) are shown in Figure 2 for the individuals that have completed the study thus far. Presented are results for the 15.8 mg/g control (i.e., usual brand cigarette) dose and the VLNCC 0.4 mg/g dose, which has the lowest addiction potential. These also represent the two doses that we are proposing to study in this renewal. Thus far, there is no evidence of sustained compensatory smoking in any population receiving VLNCCs. CPD across the two doses separates over time in all three vulnerable smoker groups; however, it does so later and overall consumption is greater among smokers with OUD. Additionally, the current effect size for differences in CPD at 12 weeks among the disadvantaged women and smokers with AD (Cohen's d=0.70 and 0.81, respectively) are



Figure 2. Total cigarettes smoked across 12-week period in three vulnerable populations.

larger than those seen in the opioid dependent population (d=0.38)consistent with and those seen at 6 weeks the general population of smokers  $(0.79^{51}).$ **Fagerstrom** dependence scores at 12 weeks are also significantly decreased

among those assigned to VLNCCs vs. the 15.8 mg/g dose in the disadvantaged women and those with AD but not in individuals with OUD. The overall greater cigarette demand and consumption exhibited by smokers with OUD serves as an important reminder of the especially persistent nature of smoking in this population.

#### 3.2. Increasing appeal of alternative non-combusted nicotine sources

These data provide promising initial evidence that smokers with concomitant other socioeconomic, substance use and psychiatric vulnerabilities will respond to RNCCs with subsequent reductions in cigarette demand and other measures of addiction potential. However, there is growing recognition of the critical importance of having appealing alternative noncombusted nicotine sources readily available if the potential of a reduced nicotine standards policy for combusted products is going to be realized. In the words of Benowitz and colleagues, "The RNCC and the emergence of non-combusted nicotine products like e-cigs should be viewed not as alternatives but as complementary components of regulatory interventions that could virtually end combusted tobacco use."52 Further, the primary conclusion of the 2014 Surgeon General's Report noted that "the promotion of noncombustible tobacco products is much more likely to provide public health benefits only in an environment where the appeal, accessibility, promotion, and use of cigarettes and other combusted products are being rapidly reduced." Our data also lead us to anticipate that smokers with OUD and perhaps other SUDs may persist in smoking even if cigarette nicotine content is reduced to very low levels. This further highlights the critical importance of having non-combusted alternative sources of nicotine readily available at reinforcing doses and in forms that enhance appeal. We know of only one report empirically examining how the presence of non-combusted products influences use of VLNCCs and that was an exploratory study of participants selected from the general smoker population.<sup>44</sup> In that study, when individuals assigned to VLNCCs opted to also use a non-combusted product, they overwhelmingly chose e-cigs over other non-combusted options (i.e., snus, NRT). This is consistent with other research modeling the substitutability of non-combusted tobacco products



for combusted cigarettes<sup>53</sup> and serves as the rationale for us focusing on e-cigs in this renewal application.

#### 3.3. E-cig use

E-cigs consist of a cartridge containing an e-liquid nicotine solution, propylene glycol (PG), vegetable glycerin (VG), flavoring, and other additives, which are heated with an atomizer that vaporizes the solution. First generation e-cigs resemble cigarettes and are disposable or rechargeable. Second generation products (and the product used in this study) often resemble pens and have refillable e-liquid reservoirs, while third generation devices have larger batteries, adjustable power delivery and replacement heating coils and wicks.<sup>54</sup> Nicotine delivery from ecigs can be comparable to those from cigarettes, depending on e-cig characteristics, nicotine content and user topography. 55-58 Toxin and carcinogen levels appear to be lower than those from cigarettes. Hecht et al. 59 reported that former smokers who had switched to e-cigs had 59-99% lower levels of 6 tobacco toxicant and carcinogen metabolites than ongoing smokers, comparable to reductions seen in smokers who had switched to nicotine lozenges.<sup>42</sup> Another study found that NNAL, a metabolite of the tobacco carcinogen NNK, was reduced by 64% in smokers who had switched to e-cigs for two weeks, as was chest tightness. 60 Initial data suggest that e-cigs may be a promising tool for supporting transition away from combusted cigarettes in smokers with OUD. 61-64 In a recent observational study with methadone- and buprenorphine-maintained smokers, 99% were familiar with e-cigs, 73% had ever tried them, and 34% were currently using e-cigs.<sup>65</sup> As in the general population, smokers with OUD reported that their reasons for e-cig use are primarily to quit or reduce smoking.65

#### 3.4. E-cig effects on smoking

E-cig use is associated with smoking reduction 66-68 and possibly quitting. In a trial using second generation e-cigs, cigarette abstinence rates were 34% after 8 weeks and 21% 6 months later, with an overall 60% reduction in CPD.69 The only published study to our knowledge on the effects of e-cigs in smokers with OUD was an uncontrolled, 6-week pilot study with 12 methadone-maintained smokers. E-cig use was associated with significant reductions in self-reported combusted cigarette use, few adverse effects, and excellent e-cig adherence (89%70). While e-cigs can reduce cigarette craving and nicotine withdrawal, 55,69,71-72 these effects are generally determined by the extent to which e-cigs are used by smokers; in turn, determinants of e-cig use include product appeal and reinforcing effects.73

#### 3.5. Importance of e-cig flavors

Over two-thirds of adult e-cig users use a flavored e-cig.<sup>5,74</sup> Flavors have been shown to substantially enhance e-cig appeal and relative reinforcing effects<sup>75-76</sup> and have been cited as a key feature affecting e-cig use among adults.<sup>5,77-78</sup> Experimental studies show that flavors increase demand for e-cigs among cigarette smokers.<sup>79-80</sup> Studies of e-cig users also highlight that flavors play an important role in their experience of the product as well as reducing cigarette consumption and craving.<sup>81-84</sup> Importantly, there is a higher prevalence of flavored tobacco use among smokers with SUDs relative to the general population.<sup>5,12,14</sup> A growing literature also suggests that opioid-dependent individuals may be especially sensitive to flavors, as activation of the mu-opioid receptor by opioid administration is associated with increased preference for sweet flavors.<sup>85-90</sup> These data suggest that combining a non-combusted nicotine source with a preferred, likely sweet, flavor may have substantial appeal and thus potential for reducing combusted cigarette use in OUD smokers.



#### 3.6 Products to be tested

#### Cigarettes to be assessed

The cigarettes to be used in this study were made under an NIH contract with production being overseen by the Research Triangle Institute (referred to as "Spectrum cigarettes"). NIH currently has approximately 10 million of these cigarettes (of varying types) for research purposes. The cigarettes selected for the study span the range of yields likely to produce the hypothesized effects, as described above. Spectrum cigarettes are not currently commercially available, although they are similar in many ways to marketed cigarettes (e.g., similar manufacturing, filter, paper, etc.).

#### E-cigarettes to be assessed

Both the JUUL and the Vuse Solo will be used and assessed in this study. While JUUL will be offered to all participants, participants that are unwilling to use JUUL will be offered the Vuse Solo. JUUL is a commercially available closed system containing two components. One component contains a lithium-ion battery (200 mAh), nichrome coil heater, silica wick, and stainless steel vapor path. The other component is the prefilled e-liquid container that also serves as the mouthpiece. Each commercially available cartridge holds approximately 0.7 mL of e-liquid containing approximately 40 mg of nicotine or 5% nicotine by weight (NBW). A lower dose containing approximately 23 mg of nicotine per cartridge or 3% NBW is also marketed but will not be used in this study. All containers contain glycerol, propylene glycol, natural oils, extracts and flavors, nicotine, benzoic acid. We will not alter the e-liquid in any way. The research staff will distribute the e-liquid containers as purchased from the manufacturer. The JUUL apparatus and 5% NBW e-liquids that will be used are legally purchasable and have been as of August 8, 2016. We will not alter them in any way.

Vuse Solo is a commercially available closed system containing two components. The power/heating device includes a 270 mAh battery, silica wick, microchips, and sensor. The other component is the prefilled e-liquid container. Each commercially available cartridge holds approximately 1 mL of liquid containing 48 mg of nicotine or 4.8% NBW. All containers contain vegetable glycerin, propylene glycol, reverse-osmosis water, glycerin, flavorings, and nicotine. The research staff will distribute the e-liquid containers as purchased from the manufacturer. The Vuse apparatus and e-liquid cartridges that will be used are legally purchasable and have been as of August 8, 2016. We will not alter them in any way.

### 3.7. Summary

Although smoking rates have declined in the overall US population, there has been little to no decline among people with OUD. A nicotine reduction strategy for combustible tobacco combined with e-cig availability may have complementary effects on smoking reductions and consequent tobacco-related health effects in this vulnerable population. This research is highly significant because it will model how the availability of e-cigs impacts the effectiveness of a reduced-nicotine policy for cigarettes in vulnerable smokers. It is responsive to the goals of the FDA in that the study conditions are designed to model real-world scenarios of possible harm reduction policies in populations that are vulnerable to smoking persistence.

### 4. Project Study Methods

This study will use a four-condition, parallel-groups research design. After a baseline period in which daily smoking rate and other baseline assessments are completed, participants will be randomly assigned to one of the following four conditions for a 16-week experimental period: (1) normal nicotine content cigarettes (NNCCs, 15.8 mg/g) alone, which serves as the control condition; (2) very low nicotine content cigarettes (VLNCCs, 0.4 mg/g) alone; (3) VLNCCs + tobacco-flavored nicotinized e-cigs (TF e-cig, 4.8 - 5.0% nicotine by weight, NBW, if they



choose to use the Vuse or JULL devise, respectively); or (4) VLNCCs + preferred-flavor nicotinized e-cigarette (PF e-cig).

# 5. Study Screening Procedures

## 5.1. Participants

Participants will be men and women, ages 21-70, who are currently receiving methadone or buprenorphine maintenance for OUD. They must report smoking ≥5 cigs/day for the past year and provide a breath CO ≥ 8ppm or a positive urine cotinine value. They must be sufficiently literate to complete research tasks, be in good physical health without serious illness or change in health in the past 3 months, must not be daily e-cigarette users, and have the technological capabilities to complete weekly face-to-face video assessments and the compatibility to use ico Smartphone Smokerlyzers for assessing breath carbon monoxide (CO) levels.. As opioid and cocaine use can directly increase smoking rates, 91-96 participants must be maintained on a stable methadone or buprenorphine dose with no regular illicit-drug abuse (<4 positive specimens) for the past month. Consent to confirm dose and drug abstinence with the participant's opioid clinic will be obtained at intake, and we will monitor any changes in dose throughout the study. These practices have been effective for confirming clinical stability in our prior smoking trials with opioid-maintained patients. 50,96-100

We will exclude those <21 years old as users below that age have legal restrictions on ability to purchase these products that can alter use patterns for reasons that do not apply to adult populations. We will exclude pregnant and nursing women and women not reporting use of contraceptives. anyone currently using nicotine replacement, bupropion or pharmacotherapies as cessation aids, those who report daily use of e-cigs in the past 30 days as they may not be compliant with the study e-cigs, and anyone intending to guit within 3 months, as participation in this study may not reduce smoking and could increase smoke and/or nicotine exposure. Those who exclusively use roll-your-own cigarettes or used other non-cigarette tobacco products (e.g., cigars, smokeless) ≥10 days in the last 30 are excluded as their use of these products may reduce the validity of our main outcome measure, total CPD (which includes study and non-study cigarettes). The following conditions are excluded as they could affect participants' abilities to complete the study: unstable medical or medication conditions (significant changes in a serious medical condition in the past 3 months, medication changes in the past 4 weeks; details provided in Protection of Human Subjects section), symptoms of psychosis or dementia, pastmonth suicidality, current (past-6 months) alcohol or SUDs other than nicotine and the OUD for which they are being treated, positive toxicology screen for illicit drugs (marijuana allowed; one re-screen opportunity), positive breath alcohol level (BAL) at screen (one re-screen opportunity). Participants who meet criteria and provide written informed consent will be enrolled into the trial.

#### 5.2. Recruitment

This study will be conducted at the University of Vermont (UVM) in Burlington, VT (primary site) and Johns Hopkins University (JHU) in Baltimore, MD. This collaboration will permit us to complete this study expeditiously, enhance sample diversity, and facilitate meaningful collaboration across multiple sites. Participants will be recruited through advertisements posted in local opioid treatment clinics, in local newspapers, on community bulletin boards, Craigslist, Facebook and word of mouth. Participants can choose to complete the pre-screening questionnaire online or by phone. At UVM, individuals recruited from online sources will be directed to a UVM-hosted recruitment website where they will have the opportunity to select which research studies interest them. They will then be redirected to a brief online screener to assess eligibility. Those who contact us by phone will be given a description of the study and asked questions to assess eligibility. The RA will read a script briefly explaining the study. Participants will be informed that this is not a smoking cessation program, and that



smoking cessation services are available in the community independent of their decision to participate in this study. If interested and eligible, participants will be asked to present for a brief 10-minute in-person medical consent visit where research staff obtain informed consent to contact participant's opioid treatment provider to confirm stability in treatment. Participants will be asked to provide a urine sample for toxicology screening. If interested and eligible following the medical consent visit, they will be invited to participate in the first portion of the screening interview. Research assistants will inform eligible participants that the screening will occur over video chat, and will assist the participant with setting up an appropriately secure video platform.

During this first portion of the screening, the participant will complete questionnaires through REDCap online while the research assistant is present over video chat or phone to deliver instructions and to answer any questions. The participant will then answer interviewer-administered questionnaires over video chat. Participants who did not yet set up their video platforms will do so with the research assistant before beginning any questionnaires. Participants will be instructed to have picture identification (e.g. driver's license) available to show the staff. If participants anticipate not having acceptable ID, staff should consult with the project coordinator or study PI. Initial study eligibility will be determined after data are collected from this visit. Participants who meet initial study eligibility will be scheduled for the second portion of the screening.

Before the second portion of the screening occurs, eligible participants will receive the equipment necessary to use for collecting physiological measurements. Participants will be asked to pick up this equipment via curbside pickup at our clinic (UVM University Health Center, UHC), which will consist of participants calling staff once they arrive at UHC and staff coming out to give participants a bag/box containing the following equipment: a Smokerlyzer; an audio jack adapter for the Smokerlyzer if necessary; a blood pressure cuff; an oximeter; a thermometer; a urinary cotinine dipstick; urine cups with attached temperature test strips; a pregnancy test strip (if applicable) and urine toxicology test strips or a saliva toxicology test. Participants (and staff) will be asked to use cloth face coverings when exchanging product. Participants may be invited to come inside to pick up this equipment if the participant is asked to wait for this exchange. All participants must pass a COVID19 screening before entering the building. If there is any waiting that needs to occur inside the building, the participant will wait inside one of our five highly ventilated smoking chambers. If there happens to be no space in the smoking chambers, the participant will be told that they can not come up to the clinic until space is available. After each use, the all of the surfaces in the smoking chambers will be cleaned with 70% or greater of alcohol solution by staff wearing a mask and gloves, as well as all of the door handles. If the participant uses the bathroom while they are in the clinic, the bathroom surfaces and handles will be wiped down after use by staff while masks and gloves are worn. Participants who are using the smoking chambers at any point in the study to wait for product or equipment exchange will remain in the chambers until a staff member comes to knock on the door to let them out. In this way, we can avoid people coming into close contact with each other in the larger room that contains the smoking chambers. A minimum of 6 feet of distance will be maintained for all staff and participants at all times. For participants who cannot come to the clinic, a commercial courier will deliver this equipment to them before the second portion of the screening.

If at any point the Smokerlyzers are not available for distribution, we will conduct the CO test curbside before or after participants are invited inside and the courier service will not be available. Research Assistants will bring down the CO monitor to the participant. While maintaining 10 feet of distance and wearing gloves, staff will explain how the CO monitor works. Once the participant is ready, staff will press the button to obtain the measurement and will set the CO monitor down and will back away 10 feet. The participant will then come to pick up the device and will blow into the monitor. After the participant completes the test, they will set down the monitor and back up 10 feet and staff will retrieve the monitor. After every use, staff will wipe down the CO monitor with disinfectant wipes and hydrogen peroxide wipes. When using the



monitor, a D-piece (a portable valve filter) must be placed into the monitor and then the single use plastic mouthpiece is placed into the D-piece. The monitor has built in SteriTouch technology to ensure optimum infection control, and the D-pieces filter out 99.9% of airborne bacteria and greater than 97% of viruses for excellent infection control. Each participant will be assigned their own D-piece to use throughout the study, and no D-piece will ever be shared among participants. Participants will gently exhale into the D-piece for the breath carbon monoxide reading. Participants will be instructed only to exhale through the device, not to inhale. D-piece technology also includes a one-way valve that prevents air from being drawn back from the monitor. D-pieces will also be wiped down after each use with disinfectant wipes and hydrogen peroxide wipes and stored in a container at the lab.

Once participants have received the necessary equipment to complete the physiological portion of the screening, the research assistant will initiate a video call with the participant. During this call, the participant will be instructed on how to use the equipment and then will be asked to use the equipment to obtain the following physiological readings: blood pressure, heart rate, oxygen saturation, temperature, and breath CO levels. Participants will also be asked to collect a urine or saliva sample during the visit. If a saliva sample is collected, the participant you will provide the saliva sample over video chat while the staff observes. If a urine sample is collected, staff will ask participant to bring this urine sample to the video screen after collection to perform a urine toxicology test and a pregnancy test (if applicable). These urine cups will have temperature strips affixed to ensure that the sample is valid. Participants who have a carbon monoxide level of less than or equal to 8 will also be asked to use the urinary cotinine dipstick to determine whether they are positive for cotinine. The participant will obtain the physiological readings and perform the tests and then will hold the results of the test up to the camera so that the research assistant can interpret and record the readings on REDCap,

UVM participants will be primarily recruited from our university opioid program, The Chittenden Center (CC). Dr. Sigmon is the Director of this clinic, which currently has 1,000 methadone- or buprenorphine-maintained patients. A survey of CC patients indicates that 88% currently smoke, which translates to approximately 880 smokers at our on-site clinic alone. Recruitment will also draw from patients receiving treatment at the office-based buprenorphine practices throughout the Burlington, VT community. JHU participants will be recruited primarily from two clinics located directly on the JHU Bayview Medical Center Campus: Addiction Treatment Services, a methadone clinic with 500 patients, and Comprehensive Care, a primary care clinic with 300 patients receiving buprenorphine. Should these resources be inadequate at any point in time, we will also recruit from two large community-based methadone programs in Baltimore with whom Dr. Stitzer has an on-going relationship as a PI of the NIDA Clinical Trials Network. Taken together, our access to opioid-maintained smokers is more than adequate to fulfill the recruitment needs of this project. Power estimations were based on the 15% dropout rate across populations in our current trials. Using an intent-to-treat approach, we require 75 randomized in each condition (300 total) to test our primary aims.

Participants will be also instructed to have handy a pack of their usual brand cigarettes, all prescription medications they are currently taking and identification (example, driver's license) during this second portion of the screening visit. If participants anticipate not having acceptable ID site staff should consult with the project coordinator or study PI.

A participant must complete his/her two-part screening session within 90 days of completing the pre-screening questionnaire. If the participant is not able to complete the two-part screening visit in that timeframe, he/she will need to complete the pre-screening questionnaire again.

#### **5.3. Informed Consent Process:**

Before beginning the informed consent process, potential participants will need to produce identification as described above. The interviewer will confirm the age and identity of the



participant. If the participant is not between the ages of 21 and 70, he/she will be dismissed without payment. During the first portion of the screening session, study information will be presented and documentation of the participant's informed consent via electronic signature on REDCap will be required prior to participating in the screening session. In order to ensure adequate informed consent, participants will be asked to read the first several lines aloud (to determine literacy) and will then be given ample time to read the consent document. If the interviewer suspects the participant is not literate, he or she will have them continue reading further to confirm. Inability to read and comprehend written study materials will result in ineligibility and the interviewer will inform the participant that they are not eligible. Only after the participant and the researcher are fully satisfied that the participant understands the purpose of the study, the confidentiality of the data, the procedures, the risks/benefits and his/her rights as a research participant will the consent form be signed and the participant undergo screening procedures.

#### 5.4. Screening Measures

Those who consent will be screened for eligibility using the following measures:

# The following physiological measures will be collected and entered directly into REDCap by the interviewer:

- 1) Expired breath carbon monoxide (CO) levels will be assessed using a Smartphone Monitor (Covita for remote collection) or a Bedfont CO monitor (for curbside collection), a reliable and valid measure of recent smoking.
  - a. <u>Urinary cotinine test strips</u> will be used to asses urinary cotinine levels if a participant's CO reading is less than or equal to 8 ppm.
- 2) A urine or saliva toxicological screen will be performed to assess the presence of illicit drugs including up to the following drugs: marijuana, cocaine, opiates, oxycodone, benzodiazepines, barbiturates, amphetamines, methadone, buprenorphine, methamphetamines, MDMA and PCP. Participants who fail the drug screen for drugs other than marijuana or their prescribed opioid medication may reschedule the interview but will need to be re-consented to ensure they have received adequate informed consent. They will be excluded if they are positive for drugs (other than marijuana or prescribed medications as determined by PI on a case-by-case basis) the second time.
- 3) <u>Urine Pregnancy Test (HCG detection)</u> will be performed for all participants.
- 4) Blood pressure and heart rate will be measured using an automated blood pressure monitor and a finger pulse oximeter to help the licensed medical professional determine final participant eligibility. Participants will be told if their blood pressure is in an abnormal range and advised to see a doctor by research staff. The research staff will also submit a medical event form for the LMP to review along with a Blood Pressure and Heart Rate Symptom Checklist form to ascertain details of the symptomatology for the LMP to review. In severe cases, the LMP may also choose to call the participant to follow-up and/or withdraw the participant from the study if necessary. All of these procedures are documented in our Blood Pressure/Heart Rate Collection: Standard Operating Procedure form which we can submit to the IRB if the Committee deems necessary.
- 5) Body temperature, respiratory rate and oxygen saturation will be added as physiological measures based on the CDC recommendations and those of Dr. David Kaminsky. https://www.cdc.gov/tobacco/basic\_information/e-cigarettes/severe-lung-disease/healthcare-providers/index.html

The following screening assessment will be administered as an interview:



1) The Mini International Neuropsychiatric Interview (MINI) 7.0<sup>70</sup>

# The following screening assessments will be administered as an interview and entered directly into REDCap by the interviewer:

- 1) The MINI Plus Modules
- 2) The MINI suicide subscale<sup>104</sup> to evaluate suicide risk.
- 3) MINI Follow-up Questionnaire (if applicable)
- 4) <u>Tobacco Use History and Exposure Questionnaire</u>, which measures variables such as smoking amount, cigarette brand, age of initiation of smoking, number of quit attempts, duration of guit attempts and duration of smoking.
- 5) Smoking Cessation Therapy Use Questionnaire
- 6) <u>Time Since Last Cigarette Questionnaire</u>
- 7) Maintenance Drug Dose Questionnaire Screening Version
- 8) <u>Medical History Questionnaire</u> to assess current diagnoses, symptoms and past health problems.
  - a. Medications will be recorded directly onto the Concomitant Medications form in REDCap.
- 9) <u>Drug Abuse Screening Test (DAST-10)</u>, which assesses quantity and frequency of alcohol and drug use (12 month and 1 month version)

# The following screening assessments will be completed by the participant directly in REDCap, except where noted otherwise:

- 1) <u>Demographic History Questionnaire</u>, which will assess age, gender, ethnicity, race, education, income, marital status, and employment history.
- 2) <u>Alcohol Use Questionnaire---based on the Alcohol Use Disorders Identification Test<sup>105</sup></u> (12 month and 1 month version)
- 3) <u>Drug Use Questionnaire---based on the Drug Abuse Screening Test<sup>106</sup> (</u>12 month and 1 month version)
- 4) Fagerström Test for Nicotine Dependence (FTND)<sup>107</sup>;
- 5) <u>Wisconsin Inventory of Smoking Dependence Motives-Brief Scale (WISDM)</u><sup>108</sup> will be administered to assess nicotine dependence severity.
- 6) Penn State Electronic Cigarette Dependence Index 109;
- 7) Smoking Stages of Change Algorithm<sup>110</sup>;
- 8) <u>Identifying Information Form</u> will include the participant's REDCap Subject Identifier, name, address (including the county of residence), email address, phone number, age, date of birth, and social security number (if applicable).
  - a. This form will be entered into the 'Identifying Information Access Database'.
    - i. Each site will have a separate 'Identifying Information Access Database'.
    - ii. Identifying information will not be shared with other sites. Each site is responsible for maintaining confidentiality of this information.
    - iii. Identifying information will be kept in a locked file cabinet (source document) and in a password protected Access Database (electronic version) separate from all other study data.
- 9) <u>Beck Depression Inventory</u> (BDI-II)<sup>68</sup>, to assess depressive symptoms.

  (This form has been updated on 1.29.20 so as to use the BDI-II. The BDI-II will be used instead of the BDI so that the data collected will be directly comparable to other projects using the BDI-II).



- 10) Overall Anxiety Severity and Impairment Scale 69(OASIS); to assess frequency and severity of anxiety symptoms.
- 11) COVID19 Symptom Questionnaire
- 12) Respiratory Symptom Questionnaire will be administered to assess respiratory health

In the event that the REDCap website is not functioning, the assessments will be administered aloud and participant answers will be recorded securely. The interviewer will enter the data into REDCap when it resumes functioning properly. This information should be recorded in the 'End of Visit Evaluation Form'.

#### 5.5. Suicidality/Mental Health Monitoring

Participants who endorse suicidal intention in the past month or a suicide attempt in the past 6 months as indicated on the BDI (score > 1 on question 9) or MINI suicide subscale (endorse question 4 and/or 5 on the MINI suicide subscale or question 6 on the MINI suicide subscale with suicide attempt in the past 6 months) or answer "yes" to question A3g on the MINI Neuropsychiatric interview and symptoms have occurred in the past two weeks will be assessed by a clinician for eligibility and possible intervention. The research staff member will contact a licensed clinician for evaluation. In the event that no clinician is available, staff will put the participant in contact with the National Suicide Prevention Lifeline at 1-800-273-8255. They will also contact the Study Coordinator and Site PI to inform them of the situation as soon as possible. Additionally, they will contact the Project Coordinator to inform her of the situation. The participant will be paid \$25 (+\$25 bonus if applicable) and provided with local mental health resources. Post enrollment, any report of suicidal ideation or attempt by a participant will be grounds for immediate withdrawal from the study.

#### 5.6. Inclusion/Exclusion Criteria

Inclusion Criteria:

- 1) Men and women ages 21-70, who are currently receiving methadone or buprenorphine maintenance treatment for opioid dependence;
- 2) Report smoking ≥ 5 cigarettes per day for the past year;
- 3) Provide an intake breath CO sample >8 ppm, (if ≤ 8 ppm, then urinary-cotinine strip must be positive);
- 4) Be without current (within the past year) serious mental disorder that would interfere with study results of completion as determined by the licensed medical professional or PI,
- 5) Be sufficiently literate to complete the research-related tasks;
- 6) Be in good physical health without serious illness or change in health or medication (not including methadone or buprenorphine dose) in the past three months as determined by the licensed medical professional at each site;
- 7) Participants must be maintained on a stable methadone or buprenorphine dose for the past month, with no evidence of regular illicit-drug abuse (<30% positive specimens in the past 30 days).
  - a. Consent to confirm dose and drug abstinence with the participant's opioid clinic will be obtained prior to screening at a medical consent visit and we will monitor any changes in dose throughout the study.
  - b. Participants must provide proof of at least three biochemical (e.g. urine, saliva) samples within the last 30 days of the date of the medical consent visit that have no evidence of illicit drug use. If they do not have three, they will be asked to provide additional samples as needed and coordinated by research staff to confirm



clinical stability. They may provide up to two samples per week with at least one full day between samples.

8) Have appropriate equipment to complete face-to-face video assessments and use ico Smartphone Smokerlyzer Monitors. For those who do not have a Smartphone, staff will explore potential alternate plans (e.g., project-provided inexpensive Android phone)

## **Exclusion Criteria:**

- 1) Exclusive use of roll-your-own cigarettes;
- 2) Planning to quit smoking in the next 30 days;
- 3) A quit attempt in the past 30 days resulting in greater than 3 days of abstinence;
- 4) Significant use of other tobacco or nicotine products within the past month (more than 9 days in the past 30).
- 5) Currently taking anticonvulsant medications including:
  - a. Phenytoin [Brand Name: Dilantin]
  - b. Carbamazepine [Brand Name: Tegretol, Carbatrol, Equetro, Epitol]
  - c. Oxcarbazepine [Brand Name: Trileptal]
  - d. Primidone [Brand Name: Mysoline]
  - e. Phenobarbital
- 6) Positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, oxycodone, buprenorphine, benzodiazepines, barbiturates, amphetamines, methamphetamines, MDMA and PCP will be grounds for exclusion.
  - a. Marijuana will be tested for but will not be an exclusionary criterion. Participants will be discouraged from smoking marijuana during the study.
  - b. Participants with valid prescriptions for opiates, benzodiazepines, barbiturates, or amphetamines will not necessarily be excluded.
  - c. Participants failing the toxicology screen will be allowed to re-screen once. These participants will need to be re-consented before being rescreened to ensure they have received adequate informed consent.
- 7) Not currently enrolled in a treatment program for opioid dependence and/or not currently stable on their methadone or buprenorphine dose,
- 8) Self-report of binge drinking alcohol (more than 9 days in the past 30 days, 4/5 drinks in a 2 hour period in females/males):
- 9) Systolic blood pressure < 90 or ≥ 160 mmHg;
  - a. Participants failing for blood pressure will be allowed to re-screen once.
- 10) Diastolic blood pressure < 50 or ≥ 100 mmHg;
  - a. Participants failing for blood pressure will be allowed to re-screen once.
- 11) Breath CO > 80 ppm;
- 12) Heart rate is greater than or equal to 115 bpm or less than 45 bpm;
  - a. Participants failing for heart rate will be allowed to re-screen once.
- 13) Currently seeking treatment for smoking cessation;
- 14) Being pregnant or nursing, or not report using an approved form of birth control if applicable determined by the Project Medical Director.
- 15) Have used nicotine replacement, bupropion or other pharmacotherapies as cessation aids in the past month (bupropion will be allowed for treatment of depression);
- 16) Current symptoms of psychosis, dementia or mania;
- 17) Suicidal ideation in the past month (score > 1 on the BDI question 9 or endorse question 4 and/or 5 on the MINI suicide subscale);



- 18) Reporting a plan or attempt to commit suicide, which is assessed on question A3g of the MINI Neuropsychiatric Interview Major Depressive Episode Module. Thoughts of suicide without an intent or plan is not an exclusion criteria;
- 19) Suicide attempt in the past 6 months (endorse question 6 on the MINI suicide subscale with suicide attempt in the past 6 months);
- 20) Participation in another research study in the past 30 days;
- 21) Daily use of e-cigarettes in the past month (defined as 6 7 days per week); or
- 22) Co-habitation with any research participant who has or is participating in the current study.
- 23) Oxygen saturation of < 90%
- 24) Reporting positive symptoms for COVID19

Individuals under age 21 are excluded because they cannot legally buy cigarettes. Those with unstable medical, psychiatric, or medication conditions (as determined by the licensed medical professional) are excluded as these symptoms could affect a participant's ability to complete the study. Examples include but are not limited to the following: angina, stroke, heart attack which occurred since phone screening, blood clots in the arms or legs for which the individual is undergoing active medical treatment, cancer requiring active chemotherapy or radiation therapy, severe shortness of breath caused by conditions such as uncontrolled asthma. COPD, or arrhythmia, active untreated infection such as pneumonia, active untreated endocrine disorder such as hyperthyroidism. We will exclude those currently seeking smoking treatment and those who plan to guit in the next 30 days, as participation in this study may not lead to reductions in smoking. We will exclude pregnant or nursing women and women of reproductive potential who are unwilling to use acceptable forms of birth control throughout the study if applicable determined by the Project Medical Director. We will also exclude anyone with current or recent alcohol or drug abuse problems as these factors could independently affect smoking behavior during the study. Individuals with baseline CO readings greater than 80 ppm, those with heart rate or blood pressure readings that are out of range (systolic: 90-159 mmHg; diastolic: 50-99 mmHg; HR: 45-114 bpm) and anyone who has attempted suicide in the past six months will be excluded from the study for safety concerns. Individuals who smoke 'roll your own' cigarettes exclusively will be excluded from the study because we will be unable to standardize their baseline smoking behavior. Individuals who have reported daily use of e-cigarettes in the past 30 days will be excluded as they may not be compliant with experimenter-provided e-cigarettes. Individuals who have recently participated in a research study will be excluded as participation may have changed their smoking patterns, which may preclude a stable smoking baseline. Because participants are required to complete portions of the protocol independently, they will need to be able to independently read and comprehend the study materials.

#### 5.7. Eligibility Determination:

The research assistant will review the entire screening assessment battery for initial eligibility determination, confirming the participant meets the above described inclusion/exclusion criteria. All eligibility criteria that are not related to physiological measurements will be assessed during the first portion of the screening visit, and all criteria related to physiological measurements will be determined during the second portion of the screening. The final eligibility of the participant will be determined by a licensed medical professional (MD, DO, NP, PA, Master's prepared RN or CRN) at each site after reviewing the Medical History Questionnaire, BDI, Mini Neuropsychiatric Interview, and the MINI suicide subscale. The licensed medical professional may meet with a participant if available and think it necessary for eligibility determination. He/she will sign off on eligibility prior to the first baseline visit. If the licensed medical professional determines the participant is not medically eligible to participate in the study, has current symptomatology that would interfere with interpretation of the data, or is unlikely to complete the study he/she will inform the research assistants who will contact the participant prior to the first



baseline visit. The licensed medical professional will not need to review the medical history forms of participants who are ineligible for other, non-medical reasons.

If a participant fails the urine or saliva toxicology screen due to a prescription medication he/she is taking, then he/she will not be automatically excluded. The interviewer will make note of this when he/she submits the forms to the licensed medical professional for final eligibility determination.

Once all the screening procedures have been completed, researchers will pay participants \$25 (+\$25 bonus if applicable) for their time as long as they pass the drug tests and meet the minimum requirements for carbon monoxide or urinary cotinine levels. Participants will be paid after the completion of the study visit. If participants are deemed ineligible at any point in the screening, the participant will be paid after determined ineligible. Marijuana will be tested for but will not be an exclusionary criterion. If a participant does not pass the drug test but has a current, valid prescription that would explain the failed test he/she will not be automatically excluded and will still receive the visit payment. Participants who meet all other eligibility criteria, sans the medical criteria, will be scheduled for the first baseline visit.

At the end of the screening session, the researcher will complete the End of Visit Evaluation Form. This will allow the researcher to make note of any problems encountered during the visit and to assess the truthfulness of the participant in regards to self-report of tobacco use.

#### 6. Study Baseline Procedures

This study will use a one-week, two-session baseline period to collect baseline individual difference measures and monitor daily usual-brand smoking behavior. At Baseline 1 or within 1 business day of the Baseline 1 visit, participants will be provided their usual brand cigarettes to smoke, equivalent to 150% of their daily smoking rate. Participants will be encouraged to come to the lab to pick up their usual brand cigarettes after they complete the questionnaires and physio for the BL1 visit. Those who cannot come to the lab will receive product via a commercial courier. A time line follow back (TLFB) will be used during the period between Baseline 1 and Baseline 2 to assess the daily cigarette use for the first 7 days the participant has product. The participant must have received their UB cigarettes from the lab before the 7-day assessment period starts, and Baseline 2 must occur at least 7 days after the participant receives their usual brand cigarettes from the lab. If the baseline period extends past seven days and if the participant has run out of product, participants will need to purchase their own usual brand cigarettes. Use of a two session baseline period will ensure stability of daily smoking reports, reduce reactivity to the daily cigarette monitoring, and reduce participant burden. During the two baseline sessions, participants will complete subjective questionnaires. Each visit will last approximately two to four hours. At the end of each baseline session, the researcher will complete the End of Visit Evaluation Form This will allow the researcher to make note of any problems encountered during the visit and to assess the truthfulness of the participant in regards to self-report of tobacco use. Participants will also be supplied with saliva test equipment and urine collection equipment during the Baseline 1 product exchange so that they can collect saliva and first void urine samples during the Baseline 2 visit.

For the Baseline 1 visit and all subsequent visits, the participant will be sent a REDCap link within 15 minutes of the start of the scheduled visit to complete all of the non-interviewer administered questionnaires. The participant will complete these questionnaires on their own but can have the research assistant present on a video call if they desire. Before beginning the physiological assessment portion of the visit over video call, the research assistant must review the participant's questionnaire responses for that visit. Participants will be compensated after the completion of the study visit and when the participant has received their new product.

At Baseline 2 and all subsequent visits, after the participant has answered the questionnaires and has completed the physiological portion of the visit over video call, participants will be asked



to come to the lab for a curbside exchange of product and biological samples. Participants will bring in their used and unused product from the previous visit as well as a first-void urine sample for assessing tobacco-related toxin exposure and a salivary sample for assessing nicotine metabolism rate on applicable visits (BL2, Week 8 and Week 16) using equipment that was provided at the previous visit. Participants will be instructed to call the RA at the office when they get to the clinicto ensure that there is enough space in the smoking chambers to house all participants while abiding by safety guidelines as detailed on page 14 of the protocol. All participants must pass a COVID19 screening before entering the building. When invited into the lab, the participant will be shown to a smoking chamber and will instructed to place their bag of product outside of the chamber. The participant will wait here while the RA processes and returns product through the randomization database. Then the RA will dispense new product and bring the bag back to the participant. When the RA deems it safe for the participant to exit the chamber, the RA will instruct the participant that they can leave. The RA will instruct the participant to observe social distancing measures during this exchange, providing clarification if necessary. If a participant forgets their first-void urine sample at the Baseline 2 visit, staff will ask participant to come back to the clinic with their first void urine sample before exchange of product occurs. If participant is unable to return to the clinic with their first void sample, staff can arrange to meet the participant off campus to pick up their urine sample and to give participant their study product. Distancing and safety measures as described above must be observed. For participants who cannot make it to UHC, special arrangements will be made to enable use of the randomization database and product return/distribution procedures to the extent possible. Each week, during - or scheduled as nearly as possible to - a virtual visit, a complete accounting of the participant's product inventory will be taken and processed remotely through the randomization database. The participant will separate product based on its type (e-cigarette or combustible inventory) and status (used/unused), and the RA will process return characteristics through the database accordingly. The RA will clarify barcode characteristics with the participant when legibility is compromised. The participant will be instructed to keep unused product in their possession, but to exchange any used product with the courier who will deliver newly dispensed replacement products within 48 hours.

Product that will be given to participants for the Baseline 2 visit cannot be given/sent to participants until 7 days have passed following completion of the Baseline 1 visit. We will need to calculate baseline smoking rate during this 7-day period and so participants cannot have access to any blinded study product or e-cigarettes before this 7-day period has ended.

#### 6.1. Visit scheduling requirements for baseline period:

Participants will be required to schedule the Baseline 1 visit within 30 days of the completion of their screening visit. If a participant still wants to be in the study after 30 days, he/she will need to be re-screened. The participant will need to be re-consented but will maintain the original REDCap Subject Identifier. The ideal target window separating Baseline 1 and Baseline 2 is between 7 and 12 days. The minimum is 7 days and the maximum is 21 days. If the participant does not complete the visit within 21 days, then he/she will not be rescheduled and will be discontinued from the study.

#### 6.2. Measures/Assessments

The following physiological measures will be collected and recorded directly into REDCap by the interviewer:

- 1) CO
- 2) Blood Pressure



- 3) Heart Rate
- 4) Body temperature
- 5) Oxygen saturation
- 6) Respiratory rate
- 7) Urine or Saliva Toxicology
- 8) Urine Pregnancy test (if applicable, to be performed every 2 weeks)

The following assessments will be administered as an interview at Baseline 1 and entered into REDCap by the interviewer at the end of the visit:

- 1) Concomitant Medications Form
- 2) Health Changes Questionnaire, which will assess any weekly health changes,
- 3) Time Since Last Cigarette Questionnaire
- 4) Maintenance Drug Dose Questionnaire

# The following Baseline 1 assessments will be completed by the participant directly in REDCap:

- 1) BDI
- 2) OASIS
- 3) Respiratory Symptom Questionnaire
- 4) COVID19 Symptom Questionnaire
- 5) <u>Wisconsin Inventory of Smoking Dependence Motives-Brief Scale (WISDM)</u> will be administered to assess nicotine dependence severity.
- 6) <u>Perceived Health Risks Rating</u><sup>112</sup>, a measure of the perceived addictive potential and other health risks associated with cigarettes;
- Perceived Stress Scale (PSS)<sup>112</sup>, assessing the degree to which life situations are perceived as stressful;
- 8) <u>Positive and Negative Affect Scales</u> (PANAS)<sup>113</sup>, a measure of changes in positive and negative mood;
- 9) Respiratory Health Questionnaire, a UVM measure of cough, shortness of breath and other respiratory symptoms;
- 10) Minnesota Nicotine Withdrawal Scale (MNWS)<sup>114</sup>, a measure of nicotine withdrawal;
- 11) Questionnaire of Smoking Urges-brief scale Usual Cigarette (QSU)<sup>115</sup>, which measures the urge to smoke;
- 12) Vaping Craving Questionnaire (VCQ) 116; which measures the urge to vape;
- 13) <u>Cigarette Evaluation Scale Usual Cigarette</u> (CES)<sup>117</sup>, which measures responses to cigarettes (e.g., reward, satisfaction);
- 14) Vaping Evaluation Scale (VES), which measures responses to vaping (e.g. reward, satisfaction)
- 15) <u>Cigarette Purchase Task Usual Brand Version</u> (CPT)<sup>118</sup>, a self-report analogue of a progressive-ratio schedule that measures the relative reinforcing efficacy of cigarettes by querying how many of that day's cigarette they would consume in a day at varying prices. This task will indicate whether prolonged VLNC cigarette use reduces cigarette demand and increases sensitivity to increases in cigarette costs;

All participants will also be asked to select their top three flavors of e-cigarette liquid from a list read to them by the RA. This question will be asked in preparation for giving flavored pods to participants who are randomized into the flavored e-cigarette condition. This information will be recorded directly into REDCap. Participants will be asked to rate these top three flavors based on either previous



experience with these flavors or to indicate how much they believe that they will like or dislike the flavors.

# Physiological measures will be collected at Baseline 2 and entered directly into REDCap by the interviewer:

- 1) CO
- 2) Blood Pressure
- 3) Heart Rate
- 4) Body temperature
- 5) Oxygen saturation
- 6) Respiratory rate
- 7) Urine or Saliva Toxicology
- 8) Urine Pregnancy (if applicable, to be performed every 2 weeks)

# The following assessments will be administered as an interview at Baseline 2 and entered directly into REDCap by the interviewer:

- 1) Concomitant Medications Form
- 2) Health Changes Questionnaire
- 3) Time Since Last Cigarette Questionnaire
- 4) Maintenance Drug Dose Questionnaire

# The following assessments will be administered at Baseline 2 and completed by the participant directly in REDCap:

- 1) BDI
- 2) OASIS
- 3) COVID19 Symptom Questionnaire
- 4) Respiratory Symptom Questionnaire
- 5) MNWS
- 6) WISDM
- 7) PANAS
- 8) QSU (usual brand)
- 9) Vaping Craving Questionnaire
- 10) CES (usual brand)
- 11) Vaping Evaluation Scale
- 12) CPT (usual brand)
- 13) E-Cigarette Flavor Rating Questionnaire
  - a. Participants will rate only the flavors that they received from staff for this visit

In the event that the REDCap website is not functioning, the assessments will be administered aloud and participant answers will be recorded securely. The interviewer will enter the data into REDCap when it resumes functioning properly. This information should be recorded in the 'End of Visit Evaluation Form'.

#### 6.3. E-cigarette Training Session (Baseline 2):

Participants assigned to an e-cig condition will be told that they will be provided with a JUUL. If a participant indicates an unwillingness to use the JUUL device, the research



assistants will offer the participant the Vuse Solo as alternative device. If the participants does not wish to use either device, he or she would be ineligible for the study.

Participants in the e-cigarette conditions will be given e-cigarette pods BEFORE the training session occurs. These pods will be either picked up at the lab (preferred) or delivered to the participant 1 to 2 days before their Baseline 2 visit occurs. Participants randomized to the e-cigarette conditions will be notified before their Baseline 2 visit (but after the 7-day period following Baseline 1) and informed of their e-cigarette condition. Participants randomized to the flavored condition will be given pods of up to three flavors of their choice. Staff will calculate how many total pods participants will be given at this time based on their smoking rate, and participants will be able to choose the proportion of each flavor that they would like to receive.

The e-cigarette training session will occur over video chat after the physiological measurements have been collected. The first 30 minutes of the training session will consist the participant being taught how to use, charge, and replace pods. Participants will first try their JUUL using the tobacco flavor. At this point, participants who are in the tobacco-only flavor condition will conclude their training session.

For all visits following Baseline 2, participants in the preferred flavor condition, participants are permitted to take up to three flavors home per week, but can choose to take less than three flavors if desired. Participants will take home their chosen pods or cartridges of up to three flavors. Participants will be able to change their flavors at only one point in the study if they desire. Participants will only be allowed to take home three flavors at one time. Participants will be given an E-cigarette instructional manual that reviews the e-cigarette training done at this visit. Participants will be encouraged to call with any device issues.

## 6.4. Interactive Voice Response System:

At the end of the first baseline visit, participants will be trained to use the Interactive Voice Response (IVR) System, which will contact participants each day throughout the study and ask about their smoking behavior as well as withdrawal symptoms the week before and after Baseline 2. We will also review the IVR adherence incentive program, which consists of \$1 per call plus a \$10 bonus for seven consecutive calls.

The IVR system is operated by TeleSage (https://telesage.com/about/). To be enrolled in the IVR system, research staff will enter the participant's initials, telephone number, subject identifier, and visit dates into the IVR TCORS website. Identifying information (initials and telephone numbers) will not be extracted as part of the data by the bioinformatics group. Please refer to TeleSage's privacy statement and HIPAA compliance form for additional information.

### **Baseline 2 biological specimens:**

1) Urine sample for smoking biomarker assessment:

Participants will be asked to provide a urine sample (first void of the day) at the second baseline session and to post-randomization weeks 8 and 16 for biomarker assessment. Biomarker analysis will provide nicotine and carcinogen exposure outcome measures and verify compliance with VLNC cigarettes. Samples will be stored at -80C. Urine samples will be analyzed for total nicotine (cotinine plus its glucuronide conjugate, a useful measure of daily nicotine exposure), the tobacco-specific nitrosamine 4-methylnitrosamineo-1-(3-pyridyl)-1-butanol (NNAL), and metabolites of 4 polycyclic aromatic hydrocarbons (PAHs), which are biomarkers of tobacco smoke carcinogens and decrease upon tobacco cessation or reduction. Anatabine is a minor alkaloid that is reduced in users of VLNC cigarettes and e-cigs. Therefore, anatabine levels in samples from those assigned to the VLNCC, VLNCC+TF e-cig and VLNCC+PF e-cig conditions should be lower than levels



from those in the NNCC condition. These analyses will be preformed by the Murphy lab at the University of Minnesota.

2) Saliva Samples for smoking biomarker assessment:

We will collect a saliva sample at the second baseline session and post-randomization weeks 8 and 16 for analysis of nicotine metabolite ratio (NMR; ratio of 3-hydroxycotininine [3 HC] to cotinine [COT]), a phenotypic marker of nicotine metabolic rate. Analyses of these samples will be performed by the Tyndale lab.

#### Biomarker shipping and storage:

Biomarkers will be shipped quarterly to the University of Vermont Laboratory for Clinical Biochemistry Research (Tracy Lab). The Tracy Lab will serve as a central repository for all biomarker specimens and will be responsible for distributing specimens to the appropriate labs on a quarterly basis. Urine samples will be analyzed and stored at the University of Minnesota Murphy Lab. The saliva samples will be analyzed and stored at the University of Toronto Tyndale Lab.

#### 7. Study Experimental Procedures

## 7.1. Experimental Period:

Participants will be seen weekly throughout the 16-week experimental period. Weeks 4, 8, 12, 16 and the abstinence visit will take approximately 2-4 hours each. All other sessions will last approximately 2 hours. If a participant has a positive urine or saliva toxicology test or is visibly intoxicated as determined by slurred speech, swaying, or stumbling, the session will be rescheduled until a negative test result is obtained and intoxication is not present. As a part of each experimental visit, participants will be asked to come to UHC for a product exchange. All participants must pass a COVID19 screening before entering the building. Participants will be instructed to contact the RA at the office when they get to the clinic to ensure that there is enough space in the smoking chambers to house all participants while abiding by safety guidelines as detailed on page 14 of the protocol. All participants must pass a COVID19 screening before entering the building. When invited into the lab, the participant will be shown to a smoking chamber and will instructed to place their bag of product outside of the chamber. The participant will wait here while the RA processes and returns product through the randomization database. Then the RA will dispense new product and bring the bag back to the participant's smoking chamber and leave it on the ground in front of the chamber. When the RA deems it safe for the participant to exit the chamber, the RA will instruct the participant that they can leave. The RA will instruct the participant to observe social distancing measures during this exchange, providing clarification if necessary. At the end of each experimental session, the researcher will complete the End of Visit Evaluation Form, which will be filed in the participant's binder. This will allow the researcher to make note of any problems encountered during the visit and to assess the truthfulness of the participant in regards to self-report of tobacco use and compliance to study procedures.

#### Visit scheduling requirements for experimental period:

The ideal scheduling window between each visit is 7 days based on the date of the Baseline 2 Visit. For additional scheduling requirements, refer to the 'Scheduling Visits SOP'. If a participant misses a visit and is unable to reschedule during the window ( $\pm$  3 days), that visit will not be 'made-up' in the future. All measures that were not completed will be considered missing data and will not be collected during future visits. If a visit mistakenly occurs outside of the designated window, this is a protocol deviation. A 'Non-Medical Event Form' will need to be completed. Additionally, each visit should occur at approximately the same time of day  $\pm$  1 hour. The interval



between the time for the participant's methadone/buprenorphine dose should also be consistent for each visit (± 1 hour).

If a participant is not able to attend his/her Week 16 visit, then it should be rescheduled even if it is outside of the scheduling window. This will be documented as a protocol deviation.

# **7.2. Experimental Visits Weeks 1, 3, 5, 7, 9, 11, 13, and 15 Procedures**

#### 7.2.A. Measures/Assessments

Physiological Measures Collected and entered directly into REDCap by the interviewer:

- 1) CO
- 2) Blood Pressure
- 3) Heart Rate
- 4) Body temperature
- 5) Oxygen saturation
- 6) Respiratory rate
- 7) Urine or Saliva Toxicology
- 8) Urine Pregnancy test (if applicable, to be performed every 2 weeks)

The following assessments will be administered as an interview and will be entered directly into REDCap by the interviewer:

- 1) Concomitant Medications
- 2) Medical Event Form, if applicable
- 3) Health Changes Questionnaire
- 4) Time Since Last Cigarette Questionnaire
- 5) Maintenance Drug Dose Questionnaire

#### The following assessments will be completed by the participant directly in REDCap:

- 1) <u>BDI</u>
- 2) OASIS
- 3) COVID19 Symptom Questionnaire
- 4) Respiratory Symptom Questionnaire
- 5) MNWS

In the event that the REDCap website is not functioning, the assessments will be administered aloud and participant answers will be recorded securely. The interviewer will enter the data into REDCap when it resumes functioning properly. This information should be recorded in the 'End of Visit Evaluation Form'.

#### 7.3. Experimental Visits Weeks 2, 4, 6, 8, 10, 12, 14, and 16 Procedures:

#### 7.3.A Measures/Assessments

Physiological measures collected and entered directly into REDCap by interviewer:

- 1) CO
- 2) Blood Pressure
- 3) Heart Rate
- 4) Body temperature



- 5) Oxygen saturation
- 6) Respiratory rate
- 7) Urine or Saliva Toxicology
- 8) Urine Pregnancy test (if applicable)

# The following assessments will be administered as an interview and will be entered directly into REDCap by the interviewer:

- 1) Concomitant Medications
- 2) Medical Event Form, if applicable
- 3) Health Changes Questionnaire
- 4) Time Since Last Cigarette Questionnaire
- 5) Maintenance Drug Dose Questionnaire

## The following assessments will be completed by the participant directly in REDCap:

- 1) BDI
- 2) OASIS
- 3) Respiratory Symptom Questionnaire
- 4) COVID19 Symptom Questionnaire
- 5) MNWS
- 6) QSU (usual brand)
- 7) QSU (study cigarette)
- 8) Vaping Craving Questionnaire
- 9) CES (usual brand)
- 10) CES (study cigarette)
- 11) Vaping Evaluation Questionnaire
- 12) PANAS
- 13) Cigarette Purchase Task Usual Brand Cigarette Version (weeks 4, 8, 12 and 16 only)
- 14) Cigarette Purchase Task Study Cigarette Version (weeks 4, 8, 12 and 16 only)
- 15) <u>Cross-price Elasticity Task<sup>120</sup>-</u> e-cigarettes and combustible cigarettes (weeks 4, 8, 12 and 16 only) (for e-cigarette experimental conditions only)
- 16) Penn State Electronic Cigarette Dependence Index (weeks 8 and 16 only)
- 17) Respiratory Health Questionnaire (weeks 8 and 16 only)
- 18) FTND (weeks 8 and 16 only)
- 19) Perceived Health Risks Questionnaire (weeks 8 and 16 only)
- 20) Smoking Stages of Change Algorithm and Contemplation Ladder (weeks 8 and 16 only)
- 21) WISDM Brief Scale
- 22) Drug Use Questionnaire 1 month version (weeks 8 and 16 only)
- 23) Perceived Stress Scale (weeks 8 and 16 only)
- 24) Alcohol Use Questionnaire 1 month version (weeks 8 and 16 only)
- 25) E-cigarette flavor rating questionnaire (weeks 4, 8, 12 and 16 only)

In the event that the REDCap website is not functioning, the assessments will be administered aloud and participant answers will be recorded securely. interviewer will enter the data into REDCap when it resumes functioning properly. This information should be recorded in the 'End of Visit Evaluation Form'.

### **Biological Samples to be collected:**

- 1) First void urine sample (Weeks 8 and 16 only)
- 2) Saliva sample (Weeks 8 and 16 only)



#### 7.4. Interactive Voice Response System:

Participants will continue to use the IVR system on a daily basis throughout the experimental period to record the number of study cigarettes smoked per day, measurement of e-cig use and use of non-study cigarettes or other tobacco products. Measurement of e-cig use will be collected by asking two questions: how many daily e-cigarette episodes occurred, where one episode consists **of around 10-15 puffs** or up to approximately 10 minutes, and what proportion of pods and/or cartridges were used per day. Participants will also be asked to log how many flavors of e-cigs they used per day. During the first week after Baseline 1, the IVR system will collect information about mood and withdrawal symptoms.

#### 7.5. Variable Incentive Program:

An incentive program has been developed with the goal of improving attendance at scheduled assessment sessions, compliance with using only study-provided tobacco products, and encouraging honest self-reports regarding all nicotine/tobacco use.

Briefly, participants will receive a total of seven tickets for each weekly visit they attend after randomization (Visits 03-18, weeks 1-16). In total, participants could earn 112 valid tickets across the 16 visits. Participants will be instructed that these tickets correspond to attendance (one ticket), honest reporting (one ticket), compliance in bringing back used and unused pods/cartridges (two tickets) and adherence to using only the assigned study product (three tickets). Participants who do not bring back all of their unused study product and used packaging will be told that they may not be eligible to earn the two compliance tickets. Participants will be further instructed that all of the tickets that they receive "could" be eligible for entry into a monthly drawing for prizes, but that only tickets that are "validated" will be eligible for prizes.

Since it is prohibitively expensive to test urine samples each week for each participant and because it is currently not feasible to detect with reasonable precision non-compliance based on biomarkers in the two higher nicotine group, we plan to only validate the attendance tickets. Hence, each participant who attends their regularly scheduled weekly session will have a total of seven validated tickets entered into the monthly drawing.

To convey the message that we may be validating honest reporting and use of only study-provided products, in a bogus pipeline of sorts, we will tell the participants that a composite assessment of the measures that we collect MAY be used to validate the amount of nicotine and tobacco products that they are using. So there is some minor deception involved, but technically we could conduct urine toxicology testing for both purposes. Hence, if the urine toxicology testing is presented as something that MAY be done for validation purposes, we feel that any deception is relatively minor. For scientific/economic reasons we are just electing to restrict validation to attendance. Nevertheless, we will debrief all participants upon the completion of the trial. We will inform them that the incentive program was based exclusively on attendance due to the relatively high cost of urine toxicology testing and other practical problems with shipping the urines for prompt testing.

Drawings will be conducted on the 1st of each month. Validation will be performed by staff who have no participant interaction and are not blind to condition. Any ticket drawn will be eligible for an incentive as the only true contingency is for attendance. There will be no mention of the basis for earning incentives (i.e., whether the ticket was for attendance, honesty, adherence). Participants will simply be informed that he or she earned an incentive from the drawing.

Each drawing will be independent (without replacement); consequently, some participants will not win a prize and others may win more than one during the study if more than one of their tickets is drawn. After confirming winners, the remaining tickets from each month will be discarded (i.e., tickets will only be entered into one drawing). The monthly prize amounts



are detailed below.

We estimate based on the 2 ½ years we think it will take to complete this study, that participants will win an average of approximately \$65 in prizes or an additional \$5.50 per week per participant.

Grand Prize (1): \$500 cash Second Prize (1): \$200 cash Third Prize (5): \$10 cash

#### 7.6. Product and Procedures Compliance Review Sessions:

At each visit, Baseline 2 through Week 16, participants will be counseled about their use of the study cigarettes and assigned e-cigarette (if applicable). Participants will be asked about any concerns or obstacles associated with use of the study cigarettes and assigned e-cigarette (if applicable). The importance of honest self-reporting will be stressed. Participants will be told that they will not be penalized for use of other nicotine or tobacco products and that it is crucial for them to report any use of these products. If difficulties are encountered, participants will be asked why they think they are experiencing difficulties (e.g., taste, withdrawal symptoms) and to problem-solve how to deal with these difficulties in order to meet the protocol requirements. Additionally, participants will be counseled about their IVR completion, visit attendance, task engagement and product accountability. Refer to the 'Product and Procedures Compliance Review Sessions SOP' for more information.

#### 7.7. Quit Attempts During the Study Protocol:

At each weekly session, we will ask each participant if s/he is currently abstaining from smoking with the intention of quitting and whether s/he is planning to quit smoking prior to his/her next scheduled visit. If a participant is currently abstaining from smoking with the intention to quit, we will encourage the participant to continue abstaining, schedule them for weekly visits, and provide them with NCI's Clearing the Air manual and local smoking cessation resources. We will give them the option of taking study product(s) home but not require that they take them, and if they do take the product(s) home we will suggest that they put the product(s) away at home so as to remove these cues from view. We will ask the participant to contact staff if they lapse and would like to receive study product(s) prior to his/her next visit. If a participant is planning to quit but has not initiated a quit attempt, we will ask if s/he has identified a quit date and if so what the date is, provide them with the Clearing the Air manual and local smoking cessation resources, provide them with the study product(s), and recommend that they put the product(s) away out of view on the quit date.

For those in a condition including e-cigarettes, we will defer to the participant's interests in continuing to use e-cigarettes as part of their quit attempt. Those who indicate that they will continue to use them will be given their same weekly supplies base on their baseline smoking rate. Those who indicate that they are planning to abstain from both combusted and non-combusted tobacco, we will honor that request. As we state above about combusted cigarettes, if participant changes his or her mind about resuming e-cigarette use, they can contact us and obtain their weekly supply.

### 7.7.A. If a participant is currently abstaining from smoking with the intention to quit:

- Encourage participant to continue abstaining from smoking
- Schedule the participant for normal weekly visits
- Provide the participant with the 'Clearing the Air' manual and local smoking cessation resources



- Give the participant the option to receive study product rather than require him/her to take the product
- If the participant choses to receive the study product have him/her sign a form acknowledging that cigarette availability could be detrimental to the quit attempt. Recommend that he/she put the product "away" at home as to avoid unwanted cues to smoke.
- If the participant chooses not to receive the study product, have him/her contact the lab if he/she lapses and would like to pick up or be mailed the study product prior to his/her next visit.

#### 7.7.B. If a participant is planning to quit smoking, but has not initiated the quit attempt:

- Ask if he/she has identified a target quit date and, if so, what that target date is
- Provide the participant with the 'Clearing the Air' manual and local smoking cessation resources
- Provide the participant with the study product as usual. Recommend that on the target date he/she put the product "away" at home as to avoid unwanted cues to smoke.

#### 7.8. Abstinence Assessment Session:

After the week 16 visit, participants will be required to attend one additional visit the following day. During this visit, participants will have been encouraged to abstain from smoking until their next scheduled visit (approximately 24 hours later). The abstinence assessment session should be scheduled no less than 18 hours and no more than 30 hours after the Week 16 visit. Abstinence will be verified by an expired breath carbon monoxide level of less than or equal to 6ppm. This session will allow us to determine whether the experimental cigarettes and e-cigarette use (for the e-cigarette conditions) have reduced the effects of abstinence on these measures relative to the control conditions. If the participant does NOT meet abstinence criteria, he/she will only receive \$20 for the visit. Those who do meet abstinence criterion will do concurrent choice session detailed below.

#### 7.8.A Participants Who Meet Criteria for Abstinence

#### 7.8.A.1 Measures/Assessments

### Physiological measures collected and entered directly into REDCap by the interviewer:

- 1) CO
- 2) Blood Pressure
- 3) Heart Rate
- 4) Body temperature
- 5) Oxygen saturation
- 6) Respiratory rate
- 7) Urine or Saliva Toxicology

# The following assessments will be administered as an interview and will be entered directly into REDCap by the interviewer:

- 1) Concomitant Medications
- 2) Medical Event Form, if applicable
- 3) Health Changes Questionnaire
- 4) Time Since Last Cigarette Questionnaire
- 5) Maintenance Drug Dose Questionnaire



#### The following assessments will be completed by the participant directly in REDCap:

- 1) <u>BDI</u>
- 2) OASIS
- 3) COVID19 Symptom Questionnaire
- 4) Respiratory Symptom Questionnaire
- 5) MNWS
- 6) PANAS
- 7) QSU-brief Usual Cigarette
- 8) QSU-brief Study Cigarette
- 9) Vaping Craving Questionnaire
- 10) Cigarette Purchase Task Usual Brand Cigarette Version
- 11) Cigarette Purchase Task Study Cigarette Version
- 12) E-cigarette Purchase Task- E-cigarette Version

In the event that the REDCap website is not functioning, the assessments will be administered aloud and participant answers will be recorded securely. The interviewer will enter the data into REDCap when it resumes functioning properly. This information should be recorded in the 'End of Visit Evaluation Form'.

#### 7.8.B. Participants Who Do Not Meet Criteria for Abstinence

#### 7.8.B.1 Measures/Assessments

Participants who do  $\underline{\text{NOT}}$  meet abstinence criteria will be required to complete the following assessments:

- 1) CO
- 2) Blood Pressure
- 3) Heart Rate
- 4) Body temperature
- 5) Oxygen saturation
- 6) Respiratory rate
- 7) Urine or Saliva Toxicology

The following assessments will be administered as an interview and entered directly into REDCap by the interviewer:

- 1) Concomitant Medications
- 2) Health Changes Questionnaire
- 3) Medical Event Form, if applicable
- 4) TLFB

The following assessments will be completed by the participant directly in REDCap:

- 1) BDI
- 2) OASIS
- 3) COVID19 Symptom Questionnaire
- 4) Respiratory Symptom Questionnaire



# 7.9. Participant Compensation:

Participants will receive \$25 for the medical consent visit. Participants will receive \$25 plus a \$25 bonus for completing each screening visit, plus an additional \$25 bonus for completing the visit on time as scheduled. Payment for the first screening session will be made upon its completion. Payment for the second session will be made regardless of enrollment as long as the participant passes the drug test and meets the minimum requirements for carbon monoxide or urinary cotinine levels. Participants who do not pass the drug test or who are visibly intoxicated as determined by slurred speech, swaying, or stumbling-will not be able to complete the visit and will be asked to take another test several days after the first positive. If they are negative for the second test, they will be eligible to participate, and if they are positive the for the second text they will be excluded. Participants will receive \$100 for each study visit from Baseline 1 to Week 16. Participants will also have a chance to earn an additional \$20 bonus for every study visit that is completed on time as scheduled starting at Week 1 and ending at Week 15. Participants can receive up to \$120.00 for the abstinence session (\$20 if participant does not achieve abstinence, \$120 if participant reaches abstinence), \$40 for biochemical verification of abstinence, and up to \$306 for completing daily IVR reports of study cigarette and other nicotine and tobacco use.. There will also be a \$150 bonus distributed at Week 16 for completing the study. Participants who do not complete the entire study will receive compensation for the sessions that they do complete. Total compensation for completing Study 3, including study visit payments, daily IVR calls and end of study bonus is \$2841. As mentioned above, participants will have a chance to earn additional incentives for compliance. honesty and attendance through urine testing. Participants will be given a debit card at the beginning of the study (during the second portion of the screening visit) and compensation for each visit will be automatically transferred to the card after they complete that visit. If debit cards are unavailable, participants will be paid via an alternate method (i.e. cash or check).

#### 7.10. End of Study:

After a participant has completed all study procedures and has been paid for participation the research assistant will read the following script and give the participant the *Clearing the Air Manual*.

"If you've reduced your smoking during this study, we encourage you to continue these reductions or even consider quitting. We would like to provide you with some resources should you decide to try to abstain from smoking (give "Clearing the Air" and hotline information). Please also feel free to consult with your physician and use any medications he/she deems appropriate. We will call you in approximately 30 days to ask about your smoking since leaving the study. There is no right answer and we know how difficult quitting can be. Please just answer honestly. The call will take less than 5 minutes. Thanks again for your participation."

The following assessments will be administered using REDCap:

#### 1) End of Study Questionnaire

#### 7.11. 30 Day Follow up Phone Call:

Participants will receive a follow-up phone call between 25 and 35 days after the abstinence assessment session to assess their smoking patterns. The phone questionnaire will last less than five minutes. The questionnaire will ask if the participant is still smoking, how much and whether he/she has attempted to quit smoking since the end of the study. Participants will receive 5 variable incentive program lottery tickets for completing the call as compensation. Those who report abstinence will be invited to complete biochemical verification and be compensated \$40 for doing so. Abstinence will be achieved by a carbon monoxide reading of 6 parts per million (ppm) or under. A urine sample may also be collected to be sent to the lab for



analysis. Additionally, any Medical Event Forms that remain open from the last session will be discussed. If the participant became pregnant during the study, this would have been recorded as a medical event. During this phone call, the research assistant will confirm her due date. This event will remain open until delivery. At that time the licensed medical professional will contact the participant to ask a few questions about the baby's health and will update the Medical Event Form.

Once a participant has completed all study procedures and all open events have been closed, the PI or Project Manager will review the participant's record and sign a form indicating study completion for that participant.

### 8.0 Study Randomization

#### **8.1 Randomization Process**

At the end of Baseline Session 2, participants will be randomized in equal probability to one of the four groups (NNCC, VLNCC, VLNCC + TF e-cig, VLNCC + PF e-cig) for a 16-week period, with stratification by site and menthol cigarette status. Participants will be randomized, using block randomization, in equal number to the dose conditions, with randomization stratified by study site and menthol status. Each site will randomize participants until the total goal of 310 participants across both sites is reached (205 at UVM and 105 at Johns Hopkins), and no effort will be made to recruit a specific number of menthol and non-menthol smokers at each site.

The lead statistician will create a randomization schedule for each of the two sites, amounting to 150% of expected enrollment at each site. The excess randomization codes will be used in the event that a site will have to enroll extra participants due to unexpectedly slow enrollment at another site. The nicotine doses will be identified by letter code and only Administrative Core personnel with no participant contact will have the link between the statistician's letter code and dose assignments. There will be no blinding of e-cigarette conditions. The Administrative Core will maintain the randomization schedule and the link between the alphabetic code and treatment assignment securely. A second sealed copy will be secured in a separate building to protect against loss related to fire or other unforeseen events.

The University of Vermont will be responsible for removing all identifying information from cigarettes received from the Research Triangle Institute (RTI), labeling each carton with a blind code, assigning product using this blind code based on the randomization schedule being provided by the UVM Biostatistics Core, and shipping cigarettes and e-cigarettes to each site as needed based on recruitment. Each site will be responsible for tracking product received and distributed to participants, collecting unused product from participants, and returning unused cigarettes and e-cigarettes to UVM. The participants, investigators and study staff will not have knowledge of which product is given to a participant or whether different participants received the same or different product.

#### **8.2 Study Product Administration**

During the experimental period, participants will be provided with a 14-day supply of research cigarettes equivalent to 150% of their daily smoking rate. Those in the e-cigarette conditions will also be provided with a 14-day supply of e-cigarettes equivalent to their daily smoking rate. This rate will be calculated at Baseline 2 and will be an average daily smoking rate based on the IVR data that reports on the usage for the first seven days following the day of the first baseline visit. This will ensure adequate availability of cigarettes in the numerous locations participants may typically keep a supply (home, work, vehicle, etc.) as well as avoid expending the entire supply if they miss a scheduled visit. Participants will be instructed to use the research cigarettes for 16 weeks, at which point they are to discontinue product use.



If there is prior knowledge a participant will be missing a visit (i.e. planned vacation, laboratory closure, etc.), then the participant will be provided with an adequate supply of cigarettes to make up for the missed visit(s). The participant will be given a 21-day supply if one visit is going to be missed and a 28-day supply if two visits are going to be missed.

#### 8.3 Guidelines for Reporting other Nicotine Product Use

Participants will be asked to refrain from use of other non-study cigarettes during the study period. If participants have to use another nicotine product, they will be told to use a non-combustible product (gum, patch, etc.). Additionally, they will be told there is not a penalty for use of non-study products, and that it is crucial for them to report any use of non-study tobacco products. Throughout the baseline and experimental periods, an Interactive Voice Response (IVR) system will be used on a daily basis to record the number of study cigarettes and non-study cigarettes used the previous day. During the baseline and first experimental week, participants will also answer daily IVR questions about their mood. Participants will be seen weekly for assessments. Brief standardized review sessions focusing on compliance with the study cigarettes and other study procedures will be provided at each visit.

# 8.4 Product Accountability:

Participants will be required to keep track of all the products provided to them. Therefore, they will be instructed to return all unused products and empty cigarette packs e-liquid pods/cartridges to the laboratory each week. Research staff will complete the 'Product Accountability Log' as they process participants' product. Any discrepancies in the product dispensed versus product returned will be discussed and recorded in the log. Research staff will weigh all opened e-cigarette pods /cartridges that the participant returns at all visits to determine how much e-liquid was used since the participant was last seen. Empty cigarette packs and e-liquid pods/cartridges will not be saved. Unused cigarette packs and e-liquid pods/cartridges will be re-distributed to the participants during Weeks 1-15. During Week 16, remaining unused cigarettes and e-cigarette pods/cartridges returned by the participants will be collected by the research staff.

Participants who report running out of cigarettes or e-liquid pods/cartridges prior to a scheduled weekly visit will be allowed to come in for an unscheduled visit to obtain more research cigarettes. To determine whether a rate change for cigarettes is necessary, we will look at the past two CO levels as compared to the Baseline 2 CO. If the CO trend is consistent with the self-report of smoking all of the allotted cigarettes then a rate increase will be granted. The participant will then receive cigarettes at a rate of 175% of their daily smoking rate. The maximum increase is 200% of their daily smoking rate. To determine whether a rate change for e-cigarettes is necessary, we will monitor the amount of e-cigarette use the participant is reporting and showing through product return along with any unscheduled visits. The investigator may grant an e-cigarette rate increase in increments of 25%. The maximum increase for e-cigarettes will be 200% of their baseline weekly e-cigarette dispensation rate.

If participants lose more than two packs of cigarettes and/or pods/cartridges and require an unscheduled visit to the laboratory to supplement their supply, they will be told the next time they lose more than two packs they will have to wait until their next scheduled appointment to receive more cigarettes.

#### 9. Study 3 Statistical Methods and Sample Size

### 9.1 Statistical Methods

Continuous outcomes will be summarized by mean, standard deviation, median and range. Categorical outcomes will be summarized by frequencies and percentages. Skewed continuous outcomes will be log- or square-root transformed as appropriate. Variables measured at each



baseline visit will be averaged and the average will be used as the baseline measurement.. As we expect conditions to be balanced on important baseline characteristics due to randomization, our primary analysis for all endpoints will not be adjusted for potential confounders. However, a secondary analysis will be completed for all outcomes adjusting for demographic characteristics (e.g., age), that we have found to be important in prior studies. Potential moderators (e.g., SSRI vs. non-SSRI antidepressant, depression vs. anxiety disorders, BMI above or below 30) will be explored by adding that term and the moderator-by-condition term to the model. We will examine age group and gender as potential moderators in a similar fashion.

Participants will be randomized in equal probability to one of the four conditions, with randomization stratified by site and menthol cigarette status. All analyses will follow the intentto-treat principle (i.e. subjects will be analyzed according to condition assignment, regardless of compliance). The Primary Aim will examine the effects of condition on total CPD (study product and non-study product). CPD will be analyzed by week (mean over all days in a seven-day period) using a mixed model to account for repeated measures from the same individual. Models will include baseline CPD as a covariate. Using a mixed model also allows us to include the effect of study site as a random effect. Additional analyses conducted using data collected at the end of the study will use orthogonal comparisons to test for a linear trend in the decrease in CPD, such that VLNCC + PF e-cig > VLNCC + TO e-cig > VLNCC > NNCC, with the largest reduction in the VLNCC + PF e-cig condition. As we expect that differences among conditions for some of the outcomes may not follow a linear pattern, we will use related planned comparisons to test for threshold effects, specifically contrasting the NNCC condition to all three VLNCC conditions, and NNCC to the two VLNC + e-cigarette conditions. Analysis of cigarette demand, smoke exposure and tobacco carcinogens (Aim 2) as well as additional outcomes, including subjective effects, will be analyzed in a similar manner. Because Exploratory Aim 3 is based on abstinence-induced effects and will be examined using data collected at a single visit at Week 17, analysis will be based on an analysis of co-variance model. In addition to the effect of condition, we will include important covariates noted above. Exploratory analyses will also be conducted combining data collected from three of the vulnerable populations (disadvantaged women of childbearing age, opioid dependent individuals, individuals with AD) to explore potential differences in effects of study condition across these populations. This will be done with the addition of the effects of population and population-by-condition terms to the models described above. Study staff will make every effort to minimize missing data, and results of our ongoing trial suggest that this will be minimal. We will examine the missing data pattern, and if it is missing at random, will use all data available, without imputation.

#### 9.2. Sample Size

Sample size was determined using NQuery Advisor based on hypothesis tests related to Aim 1 to detect a significant difference between conditions on total CPD. The primary statistical approach will be repeated measures ANOVAs but required sample sizes were calculated

focusing on expected outcomes at Week 16. This estimate is intentionally conservative and calculated based on one outcome at one time point; however, given the repeated measures nature of our data, we will have correlated observations within subjects and thus will achieve the stated power to detect differences of even lesser magnitude. Estimates are based on preliminary results from our current trial and from the Donny et al.<sup>41</sup> study of VLNCCs and NNCCs. The between-group effect size is defined as the difference of study condition means divided by the common standard deviation. A sample size of 75 participants per condition will

| Outcome | Observed<br>between-<br>group ES (15.8<br>vs. 0.4 mg/g) |
|-----------|---------------------------------------------------------|
| CPD | 0.38 |
| Craving | 0.74 |
| FTND | 0.14 |
| Breath CO | 0.06 |

provide 80% power to detect an effect size of 0.50 for all pair-wise comparisons, with a two-


sided type 1 error rate of 0.05. While this is larger than the effect size in our ongoing trial, we assume that the addition of e-cigs to the VLNCCs will decrease CPD from that seen with VLNCCs alone. Thus, while we recognize that we may have insufficient power to detect differences between the VLNCC and NNCC alone conditions, we expect a larger effect size when comparing the NNCC and either of the VLNCC + e-cig conditions. This sample size also provides greater than 95% power to detect a linear dose-response effect across conditions. Because we have relied only on outcomes at Week 16, our proposed sample sizes are somewhat conservative, but we believe this is appropriate given that the effects of VLNCCs in this population, particularly in combination with e-cigs, are unknown. The sample size assumes a 15% loss to follow-up, consistent with our experience in the current study. We will increase our overall sample size to 310 in order to allow pilot testing with 10 participants..

# 10. Potential Risks of Participation

# 10.1 Risks of Participation

- 1) <u>Survey Questionnaires.</u> Surveys include questions about participants' medical and psychiatric histories, drug and alcohol use and history, breath tests for cigarette and alcohol use, urine or salivary tests of illicit drug use and pregnancy, and questionnaires about your mood. Answering these personal questions can make participants uncomfortable. If a participant reports thoughts of killing themselves or other indicators of suicidality, a study clinician will come to talk to the participant. The participant may also request to see a study clinician if he or she is in discomfort and would like help and/or referrals for mental health resources.
- 2) <u>Breach of Confidentiality</u>: The risk of the interview is loss of privacy if other people find out the results.
- 3) <u>Undue Influence</u>: Undue influence is a possible risk due to monetary compensation for participating in these studies. The likelihood of this risk is low because the compensation is commensurate with the amount of time and effort required for these studies.
- 4) <u>Drug Testing</u>: A breach of confidentiality could occur and other people could learn of the participant's drug use.
- 5) Obtaining Blood Pressure and Heart Rate. The blood pressure cuff may cause minimal discomfort. In obtaining blood pressure we may find a participant to have abnormal blood pressure and/or heart rate. If participant's blood pressure is abnormal, we will inform the participant of this, and participant may be advised to see a doctor, and may also be contacted by our study doctor. Also, smoking and nicotine can affect the cardiovascular system, which may result in changes in blood pressure and/or heart rate.
- 6) <u>Smoking Cigarettes</u>: All cigarettes are detrimental to a person's health and can lead to significant medical problems including:
  - a. Cardiovascular Diseases: Coronary heart disease, heart attack, stroke, peripheral vascular disease, reduced blood circulation, abdominal aortic aneurysm
  - b. Respiratory Diseases: Emphysema, bronchitis, and chronic airway obstruction
  - c. Cancers: Cancer of the lung, bladder, cervix, esophagus, kidney, larynx, mouth, pancreas, throat, and stomach; leukemia
  - d. Metabolic Diseases: Type 2 Diabetes



- e. Other Health Risks Associated with Smoking: Including but not limited to infertility, lower bone density in postmenopausal women, and hip fracture in women
- f. Death
- 7) Smoking Study Cigarettes. All cigarettes are harmful to a person's health and can lead to cardiovascular (heart) disease, respiratory (lung) disease, cancer and other health problems. In addition to the above medical problems, participants may experience some minor negative health effects such as headaches. Participants may also experience smoking withdrawal symptoms, which are listed below. In addition, due to the altered nicotine levels, there could be a change in a participant's use of cigarettes including the manner in which he or she inhales the smoke. Smoking the study cigarette does not necessarily provide any less risk than the participant's usual brand of cigarette and could pose increased health risks.
- 8) Using Study E-cigarettes. E-cigarettes are devices that heat nicotine to produce an aerosol. The health effects of e-cigarettes are still unclear, but appear to be less than that for tobacco cigarettes. Most e-cigarette users have lower nicotine levels than when they smoked regular cigarettes. Some e-cigarette users, especially those who use both e-cigarettes and regular tobacco cigarettes as well as youth and young adults, can have increased nicotine levels. In some rare cases, these use patterns have been associated with seizures. Whether this would occur with the concurrent use of very low nicotine cigarettes is unclear. E-cigarettes users very often maintain addiction to nicotine, but this addiction appears to be somewhat less than that from tobacco cigarettes. Abruptly quitting e-cigarettes could cause withdrawal symptoms similar to those from quitting tobacco cigarettes (see below) but slightly less severe. The most common side effects include dry mouth, irritation of the throat and mouth, and mild cough. The JUUL and Vuse e-cigarettes we will be providing have not been well-studied but appear to be of similar risk to other e-cigarettes. Participants may have heard that e-cigarettes, or "vapes," can explode and seriously injure people. Study staff should instruct participants that although they appear rare, these explosions are dangerous. The exact causes of these incidents are not yet clear, but some evidence suggests that battery-related issues may lead to vape explosions. In order to prevent e-cigarette related injuries, instruct participants to keep their e-cig away from other metal objects, never charge the e-cig with a phone or tablet charger, don't charge the e-cig overnight or leave it charging unattended, and to stop using the e-cig if the batteries get damaged or wet. The participant will be instructed to always keep e-cig liquid out of kids' and pets' reach and sight after use. If the study staff learns about additional risks of e-cigarettes during the study, participants will be informed of these risks.
- 9) Mood and Psychiatric Symptom Changes. Participants may experience smoking withdrawal symptoms during this study. These symptoms can include anger, anxiousness, craving for a cigarette, depressed mood, difficulty concentrating, frustration, increased appetite, impatience/impulsivity, irritability, restlessness, sleep problems, and weight gain. These feelings can be uncomfortable and can last a couple of weeks, but usually are of minimal risk. In addition, if participants have a past history of anxiety, depression, or alcoholism, it is possible withdrawal could cause substantial increases in depression and anxiety symptoms, but this appears to be rare. At each visit, study staff will ask participants how they feel. If either study staff or the participant thinks that being in this study is putting the participant's mental health at risk, staff may have the participant meet with an on-site clinician and/or stop participating in the study.



Further, if a participant report thoughts of killing oneself or other indicators of suicidality, a study clinician will come to talk to the participant. Participants may also request to see a study clinician if he or she is in discomfort and would like help and/or referrals for mental health resources.

- 10) <u>Returning to Regular Smoking:</u> It is possible that if participants return to smoking their usual brand of cigarette at the end of the study they may experience mild and transient nausea, dizziness, and lightheadedness.
- 25) Risk to Fetus. To avoid risks to a fetus, it is important that participants are not pregnant during this study. Avoiding sexual activity is the only certain method to prevent pregnancy. However, if participants choose to be sexually active, participants should be using approved forms of birth control if applicable determined by the Project Medical Director, including but not limited to prescribed birth control pills, patch, ring, injections, implants or intrauterine device (IUD) or an appropriate "double barrier" method.. If you choose to be sexually active during this study, pregnancy could still result even with the use of these birth control methods.

# **10.2** Avoiding Risks to Fetus:

If participants choose to be sexually active, they should use an appropriate "double barrier" method of birth control (such as female use of a diaphragm, or contraceptive sponge, in addition to male use of a condom) or the female should be using prescribed "birth control" pills, patch, ring, injections, implants or intrauterine device (IUD) if applicable determined by the Project Medical Director. If a participant endorses a "double barrier" method, our medical professional will speak to the participant to confirm which methods will be used during the duration of the study. Participants will be tested for pregnancy every two weeks beginning at screening through the last study visit. If a participant becomes pregnant during the study, she will be withdrawn from the study. Approximately 30 days after being withdrawn or having a positive pregnancy test at the last study visit, the research staff will call the participant to confirm her due date. The licensed medical professional will follow-up with the participant after delivery to ask questions about the baby's health.

## 10.3 Expected benefits of participation:

There are no benefits from participating in the study. The information obtained from this study may ultimately help the Food and Drug Administration decide how best to regulate nicotine and tobacco products with the goal of improving public health.

## 11. Protection Against Risk

#### 11.1 Data Collection Protections

Research data without identifiers will be maintained in a locked file cabinet and on password-protected computers in the research staff workplace, with only code numbers identifying subjects. Study consent forms and the linkage between the participants' names and codes will be stored in a locked file cabinet inside a locked office. Interviews with participants will be conducted in private rooms. Urine or saliva samples for drug and pregnancy tests and tobacco exposure biomarkers will be obtained in a private bathroom within the laboratory suite. Subjective measures will be administered electronically. The biostatistics and data-management



team will provide consistent data-management practices for all data in the Center. Using REDCap, which is housed on the University of Vermont Medical Center's HIPAA-compliant computing system, will maximize validity and reliability of data. REDCap is a secure, web-based system that accommodates local and remote data collection by each project team, and allows for data entry work-flow monitoring and data quality control monitoring by biometry staff. The RedCap database for this project will be hosted on the UVMCOM servers. In addition, data will be collected from participants on a daily basis using an interactive voice recognition system (IVR) developed and hosted by TeleSage Inc (www.telesage.com, Chapel Hill, NC). TeleSage is a company with expertise on gathering patient-centered outcomes tracking data for mental health clinical and research institutions. TeleSage has developed and hosted behavioral health-related research software systems using IVR and Web-based technologies and is leader in behavioral health outcomes tracking technologies. For data integrity, data entry windows will follow the structure of paper forms as much as possible to allow for ease of entry, and will use predefined choices to minimize errors when possible. Data quality monitoring will be facilitated with periodic down loads and analysis using a variety of common statistical program format such as SAS, Stata, R, and SPSS. Quality control procedures will be conducted for all data collected, including analysis of missing data and logic checks for out of range and other anomalous values. This secure electronic data gathering and transmission plan, overseen by the experienced biostatistical team, will minimize opportunities for breaches of confidentiality. Biological samples for nicotine and carcinogen biomarker analysis will be marked with participant ID, stored in the locked laboratory suite, and sent to a laboratory for analysis on a quarterly basis.

All information collected as part of this study will be accessible only to research staff. No information will be shared with participants' clinicians unless the participant requests this in writing. All investigators and staff have undergone (and any new staff will undergo) human subjects' ethics training as required by UVM and are fully conversant with relevant ethical principals around confidentiality. Assessments, consenting and study procedures will be closely supervised by the PI.

The sponsors (NIDA/FDA) as well as the Institutional Review Board and regulatory authorities could be granted direct access to original medical and research records for verification of clinical trial procedures and/or data. If this is required, it will be done under conditions that will protect privacy to the fullest extent possible consistent with laws relating to public disclosure of information and the law-enforcement responsibilities of the agency.

# 11.2 Data Storage:

Data will be stored locally at each site. Long-term storage of all study data, for at least 7 years after study completion, will be at the University of Vermont.

# 12. Adverse Events

The research assistant will ask about adverse events at each session, using a form that assesses the nature, severity, duration, action taken, and outcome of study-related adverse events. AEs will be captured from the time of first study cigarette. Participants will be given contact cards to inform us of events that occur between study contacts. Any AE that remains open will be reviewed and closed at an interview conducted 30 days after the study completion date (completers) or when the study should have ended had the participant completed the study (dropouts and those withdrawn by investigator).

All procedures will be monitored to ensure that they conform to the approved protocol. In addition, monitoring will be done of all unforeseen circumstances that might arise and affect safety; of all reports of serious adverse events as defined in 38 CFR 46 (death, new or prolonged hospitalization, persistent or significant disability/incapacity); of other significant



adverse events (adverse events that lead to drop out by the participant or termination by the investigator); of unexpected adverse events resulting from the study, and of expected adverse events

Any SAE will be brought to the attention of the site PIs as soon as possible and not longer than 24 hours. Any AE or SAE that is both unexpected and related to study participation will be reported to the IRB within 7 days of the event. The local IRB will make a determination as to whether additional reporting requirements are needed. IRB actions will be reported to the funding agency by the PIs no less than annually and more frequently as recommended by the local IRB. Any SAEs will be summarized in the yearly Progress Reports to the funding agency, including a review of frequency and severity. All SAEs will be followed through ongoing consultation with the physician caring for the patient until they resolve, result in death, or stabilize and are not expected to improve. The study staff will be in close contact with participants and health care providers throughout the study to monitor for potential unanticipated problems. Any unanticipated problems will be discussed at the weekly research staff meetings and reported as required to the local IRB.

# 13. Withdrawal or Monitoring of Participants

# For the participant's protection, participants will be withdrawn immediately from the study if any of the following occur:

- 1) <u>Cardiovascular disease (CVD) event</u>: Typically includes MI (heart attack), PTCA (angioplasty/stenting), bypass surgery, stroke, peripheral vascular disease (arterial blockages in arms or legs leading to procedure or surgery). Less common CVD problems would be new cardiac arrhythmias (e.g., new atrial fibrillation) or new valvular disease (e.g., mitral or aortic regurgitation).
- 2) <u>DVT/PE</u> (deep vein thrombosis/pulmonary embolism, i.e., blood clots in the venous system).
- 3) <u>Suicide Attempt</u>: A participant will be withdrawn if he/she attempts suicide at any time during participation in the study.
- 4) <u>Psychiatric Hospitalization</u>: A participant will be withdrawn if he/she is hospitalized for psychiatric reasons at any time during participation in the study.
- 5) Pregnancy: If participant indicates she is pregnant or has a positive pregnancy test at any time during the study, she will be withdrawn from the study, and this event will remain open until delivery. At that time the licensed medical professional will contact the participant to ask a few questions about the baby's health and will update the open 'Medical Event Form'. A positive pregnancy test at Week 16 will trigger a 'Medical Event Form' to be completed but will not result in withdrawal since she is no longer receiving study product.
- 6) Expired breath carbon monoxide increase: A participant will be withdrawn from the study if the average of two consecutive CO readings during the same visit is 100 ppm or greater.
- 7) Marked increase in smoking: A participant will be withdrawn from the study if he/she meets **BOTH** of the following criteria for two consecutive weeks
  - a. Cigarette per day increase: The average CPD increases by more than 100% from the average CPD during baseline.
  - b. Expired breath carbon monoxide increase: If the average of two consecutive CO measurements in the same visit is
    - i. CO is greater than 50 ppm if CO at Baseline 1 is <20 ppm.



- ii. CO is greater than 60 ppm if CO at Baseline 1 is 20 34 ppm.
- iii. CO is greater than 70 ppm if CO at Baseline 1 is 35 49 ppm.
- iv. CO is greater than 80 ppm if CO at Baseline 1 is 50 64 ppm.
- v. CO is greater than 90 ppm if CO at Baseline 1 is 65 80 ppm.
- c. Note: If the second consecutive visit is the last study visit, then the participant would not be withdrawn from the study.
- 8) <u>If a participant is discharged from or discontinues his or her methadone or buprenorphine treatment</u>, they will be discontinued from the study.

# The following will be monitored and can lead to the participant being withdrawn by the PI or Licensed Medical Professional:

- 1) <u>Cigarettes per day increase</u>: Continued participation will be evaluated by the site PI if the average number of cigarettes per day (CPD) increases by more than 100% from the average CPD during baseline as determined by CPD at Baseline 2.
- 2) <u>Blood pressure (BP) or heart rate (HR) changes</u>: If any of the following occur postenrollment: 1) BP is at or above 160/100 or below 90/50, or 2) HR is at or above 115 bpm or below 45 bpm a manual blood pressure and heart rate measurement will be taken after 10 minutes have passed. If the manual reading is still out of range, a 'Blood Pressure and Heart Rate Symptom Checklist' and 'Medical Event Form' will be completed, and the participant will be monitored by the medical professional.
- 3) Expired breath Carbon Monoxide increase: If the average of two consecutive CO measurements meets the criteria below then the 'Medical Event Form' will be completed and the participant will be monitored by the medical professional.
  - a. CO is greater than 50 ppm if CO at Baseline 1 is <20 ppm.
  - b. CO is greater than 60 ppm if CO at Baseline 1 is 20 34 ppm.
  - c. CO is greater than 70 ppm if CO at Baseline 1 is 35 49 ppm.
  - d. CO is greater than 80 ppm if CO at Baseline 1 is 50 64 ppm.
  - e. CO is greater than 90 ppm if CO at Baseline 1 is 65 80 ppm.
- 4) <u>Any hospitalization or debilitation</u> in which participation in the study could be detrimental to the recovery process. This will be self-reported by the participant and will be reviewed by the site PI and medical professional to determine whether continued participation in the study is appropriate.
- 5) If a participant is behaving in an inappropriate or threatening manner, admits to lying about eligibility criteria, is participating in other smoking research studies that could affect the primary outcome measures, etc., then the PI can withdraw him/her from the study at the PI's discretion.
- 6) If a participant fails to attend regularly scheduled research assessment visits or comply with the research procedures or schedule, then the PI can withdraw him/her from the study at the PI's discretion.
- 7) Increase in psychiatric symptoms: Exacerbation in symptoms noted during the study (i.e., change in BDI category from mild to moderate or moderate to severe) will trigger review by the study's licensed medical professional. The PI will withdraw the participant upon the licensed medical professional's recommendation.

## 14. Data Safety Monitoring Board



A Data and Safety Monitoring Board (DSMB) has been established to monitor safety outcomes and will be comprised of four members. The DSMB will be chaired by Kevin Delucchi, PhD., Professor in Residence of Biostatistics in Psychiatry at the University of California San Francisco and Director of the Quantitative Core of the San Francisco Treatment Research Center; Eden Evins, MD, MPH., Cox Family Professor of Psychiatry at Harvard Medical School and Director of Center for Addiction Medicine at Massachusetts General Hospital; Ari Kirshenbaum, Ph.D., Professor of Psychology at Saint Michael's College who he teaches courses in psychopharmacology and neuroscience, and currently has grants from NIH and NSF for work in human behavioral pharmacology and his grant-funded work focuses on cognitive and behavioral responses to nicotine and cannabinoids; and Elisabeth Johnson, Ph.D., who has over twenty years of clinical experience in women's health and pediatrics, including caring for women with substance use disorders.

#### **Conflict of Interest**

None of the board members will be otherwise affiliated with the center and each member will complete a conflict of interest disclosure form prior to each meeting. Ad hoc specialists may be invited to participate as non-voting members at any time if additional expertise is desired.

# **Monitoring Activities and Frequency of Meetings**

The DSMB will set their own agenda and decisions about monitoring; e.g. how frequently to monitor, what threshold requires changes to protocol or stopping the study, and whether to view raw or analyzed data. The DSMB will be given FDA and EMEA guidelines for DSMBs and recent reviews on DSMBs. A brief report will be generated from each meeting for the study record and forwarded to each of the study site's Institutional Review Boards (IRB) and NIDA's Program Officer with the progress report. The DSMB will be available to convene outside of the regular meetings, if necessary. If concerns should arise regarding a particular subject, or any troublesome trends in the experiences of participants, they will make appropriate recommendations for changes in protocol, as needed. The project investigators will continue to examine safety data, blind to study condition, in case they wish to make study modifications. Before modifications are made, they will inform the DSMB and request their comments.

# Communication Plan to IRB, NIDA, and FDA (if applicable)

All IRBs, the FDA and the NIDA's Program Officer will be informed of any significant action taken as a result of the Data and Monitoring Board's findings. Study Participants will be informed of any changes in risk.

### **Protection of Confidentiality**

For DSMB meetings only de-identified data, including blinded study site and condition type, will be provided to the board. All data and discussion during the meeting will be confidential.

# 15. Investigational Tobacco Product

The University of Vermont Center on Tobacco Regulatory Science will complete an Investigational Tobacco Product (ITP) application with the FDA to cover the experimental cigarettes being used in this study. This application encompasses both Project 2 sites.

# 16. Certificate of Confidentiality



To help protect the participant's privacy, Dr. Stephen Higgins, PhD, will obtain a Certificate of Confidentiality from the national Institute on Drug Abuse. With this certificate, the researchers cannot be forced to disclose information that may identify the participants, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify the participants, except as explained below. The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the Federal Food and Drug Administration (FDA).

The Certificate of Confidentiality does not prevent the participant or a member of their family from voluntarily releasing information about themselves and their involvement in the research. If an insurer, employer or other person obtains the participant's written consent to receive research information, then the researcher may not use the Certificate to withhold that information.

The Certificate of Confidentiality does not prevent the researchers from disclosing voluntarily, without consent, information that would identify the individual as a participant of the research project in instances such as evidence of child abuse or a participant's threatened violence to self or others.

#### 17. Outcome Variables

# **Primary Endpoints for Study 3:**

- 1) Cigarette Smoked per Day (CPD)
- 2) Nicotine Dependence Severity

# Secondary Endpoints for Study 3:

- 1) Measures of adherence: non-study cigarette use, drop-out rate
- 2) Measures of psychiatric symptoms: BDI, OASIS
- 3) Measures of discomfort/dysfunction: MNWS, QSU
- 4) Measures of other health-related behaviors: breath alcohol, urine or salivary drug screen, TLFB-drug use, Alcohol Use Questionnaire, Drug Use Questionnaire, weight
- 5) Measures of nicotine/tobacco dependence: FTND, WISDM
- 6) Measures of tobacco exposure: CO, total nicotine equivalents, NNN, NNAL, minor alkaloids
- Measures of intention to quit: Stages of Change, Contemplation Ladder
- 8) Measures of compensatory smoking: puff topography, filter analysis
- 9) Measures of other tobacco use: TLFB-other tobacco
- 10) Measures of cigarette characteristics: CES, Cigarette Purchase Task
- 11) Measures of cardiovascular function: heart rate, blood pressure, urine 11-dehydroTXB2
- 12) Measures of perceived risk: Perceived Health Risk Questionnaire
- 13) Safety outcome variables: Adverse Events (AEs), Serious Adverse Events (SAEs)



### 18. References

- 1. U.S. Department of Health and Human Services. *The Health Consequences of Smoking—50 Years of Progress: A Report of the Surgeon General*. Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health, Atlanta GA; 2014.
- 2. Lasser K, Boyd JW, Woolhandler S, Himmelstein DU, McCormick D, Bor DH. Smoking and mental illness: A population-based prevalence study. *JAMA*. 2000;284(20):2606-2610.
- 3. Lawrence D, Mitrou F, Zubrick SR. Smoking and mental illness: results from population surveys in Australia and the United States. *BMC Public Health*. 2009;9:285. doi:10.1186/1471-2458-9-285.
- 4. Schroeder SA. American health improvement depends upon addressing class disparities. Prev Med. 2016; 92:6-15. Doi: 10.1016/jypmed.2016.02.024.
- 5. Villanti AC, Johnson AL, Ambrose BK, et al. Flavored Tobacco Product Use in Youth



- and Adults: Findings From the First Wave of the PATH Study (2013-2014). *Am J Prev Med*. March 2017. doi:10.1016/j.amepre.2017.01.026.
- 6 .Conway KP, Green VR, Kasza KA, et al. Co-occurrence of tobacco product use, substance use, and mental health problems among adults: Findings from Wave 1 (2013-2014) of the Population Assessment of Tobacco and Health (PATH) Study. *Drug Alcohol Depend*. 2017;177:104-111. doi:10.1016/j.drugalcdep.2017.03.032.
- 7. Engström A, Adamsson C, Allebeck P, Rydberg U. Mortality in patients with substance abuse: a follow-up in Stockholm County, 1973-1984. *Int J Addict*. 1991;26(1):91-106.
- 8. Grinshpoon A, Barchana M, Lipshitz I, Rosca P, Weizman A, Ponizovsky AM. Methadone maintenance and cancer risk: an Israeli case registry study. *Drug Alcohol Depend*. 2011;119(1-2):88-92. doi:10.1016/j.drugalcdep.2011.05.028.
- Hser YI, McCarthy WJ, Anglin MD. Tobacco use as a distal predictor of mortality among long-term narcotics addicts. *Prev Med*. 1994;23(1):61-69. doi:10.1006/pmed.1994.1009.
- Hurt RD, Offord KP, Croghan IT, et al. Mortality following inpatient addictions treatment. Role of tobacco use in a community-based cohort. *JAMA*. 1996;275(14):1097-1103.
- 11. Jamal A, King BA, Neff LJ, Whitmill J, Babb SD, Graffunder CM. Current cigarette smoking among adults United States, 2005-2015. *MMWR Morb Mortal Wkly Rep.* 2016;65(44):1205-1211. doi:10.15585/mmwr.mm6544a2.
- 12. Clemmey P, Brooner R, Chutuape MA, Kidorf M, Stitzer M. Smoking habits and attitudes in a methadone maintenance treatment population. *Drug Alcohol Depend*. 1997;44(2-3):123-132.
- 13. Guydish J, Passalacqua E, Tajima B, Chan M, Chun J, Bostrom A. Smoking prevalence in addiction treatment: a review. *Nicotine Tob Res.* 2011;13(6):401-411. doi:10.1093/ntr/ntr048.
- Haas AL, Sorensen JL, Hall SM, et al. Cigarette smoking in opioid-using patients presenting for hospital-based medical services. *Am J Addict*. 2008;17(1):65-69. doi:10.1080/10550490701756112.
- 15. Mutschler NH, Stephen BJ, Teoh SK, Mendelson JH, Mello NK. An inpatient study of the effects of buprenorphine on cigarette smoking in men concurrently dependent on cocaine and opioids. *Nicotine Tob Res.* 2002;4(2):223-228. doi:10.1080/14622200210124012.
- 16. Nahvi S, Richter K, Li X, Modali L, Arnsten J. Cigarette smoking and interest in



- quitting in methadone maintenance patients. *Addict Behav.* 2006;31(11):2127-2134. doi:10.1016/j.addbeh.2006.01.006.
- 17. Richter KP, Gibson CA, Ahluwalia JS, Schmelzle KH. Tobacco use and quit attempts among methadone maintenance clients. *Am J Public Health*. 2001;91(2):296-299.
- 18. Parker M, Streck JM, Sigmon SC. Prevalence and severity of nicotine dependence in opioid-dependent vs. general population using national data. In preparation.
- 19. Clarke JG, Stein MD, McGarry KA, Gogineni A. Interest in smoking cessation among injection drug users. *Am J Addict*. 2001;10(2):159-166.
- Dunn KE, Sigmon SC, Reimann E, Heil SH, Higgins ST. Effects of smoking cessation on illicit drug use among opioid maintenance patients: A pilot study. *J Drug Issues*. 2009;39(2):313-328.
- 21. Frosch DL, Shoptaw S, Jarvik ME, Rawson RA, Ling W. Interest in smoking cessation among methadone maintained outpatients. *J Addict Dis.* 1998;17(2):9-19. doi:10.1300/J069v17n02 02.
- 22. Kozlowski LT, Skinner W, Kent C, Pope MA. Prospects for smoking treatment in individuals seeking treatment for alcohol and other drug problems. *Addict Behav*. 1989;14(3):273-278.
- 23. Sees KL, Clark HW. When to begin smoking cessation in substance abusers. *J Subst Abuse Treat*. 1993;10(2):189-195.
- 24. Nahvi S, Ning Y, Segal KS, Richter KP, Arnsten JH. Varenicline efficacy and safety among methadone maintained smokers: a randomized placebo-controlled trial. *Addiction*. 2014;109(9):1554-1563. doi:10.1111/add.12631.
- 25. Okoli CTC, Khara M, Procyshyn RM, Johnson JL, Barr AM, Greaves L. Smoking cessation interventions among individuals in methadone maintenance: a brief review. *J Subst Abuse Treat*. 2010;38(2):191-199. doi:10.1016/j.jsat.2009.10.001.
- 26. Poling J, Rounsaville B, Gonsai K, Severino K, Sofuoglu M. The safety and efficacy of varenicline in cocaine using smokers maintained on methadone: a pilot study. *Am J Addict*. 2010;19(5):401-408. doi:10.1111/j.1521-0391.2010.00066.x.
- 27. Reid MS, Fallon B, Sonne S, et al. Smoking cessation treatment in community-based substance abuse rehabilitation programs. *J Subst Abuse Treat*. 2008;35(1):68-77. doi:10.1016/j.jsat.2007.08.010.
- 28. Richter KP, McCool RM, Catley D, Hall M, Ahluwalia JS. Dual pharmacotherapy and motivational interviewing for tobacco dependence among drug treatment



- patients. J Addict Dis. 2005;24(4):79-90.
- Miller ME, Sigmon SC. Are Pharmacotherapies Ineffective in Opioid-Dependent Smokers? Reflections on the Scientific Literature and Future Directions. *Nicotine Tob Res*. 2015;17(8):955-959. doi:10.1093/ntr/ntv030.
- 30. Substance Abuse and Mental Health Services Administration (SAMHSA). *Results from the 2012 National Survey on Drug Use and Health: Summary of National Findings*, NSDUH Series H-46, HHS Publication No. (SMA) 13-4795. Rockville, MD: Substance Abuse and Mental Health Services Administration; 2013.
- 31. Substance Abuse and Mental Health Services Administration (SAMHSA). National Survey of Substance Abuse Treatment Services (N-SSATS): 2012. Data on Substance Abuse Treatment Facilities. BHSIS Series S-66, HHS Publication No. (SMA) 14-4809. Rockville, MD: Substance Abuse and Mental Health Services Administration; 2013.
- 32. Benowitz NL, Henningfield JE. Establishing a nicotine threshold for addiction. The implications for tobacco regulation. *N Engl J Med*. 1994;331(2):123-125. doi:10.1056/NEJM199407143310212.
- 33. Benowitz NL, Henningfield JE. Reducing the nicotine content to make cigarettes less addictive. *Tob Control*. 2013;22 Suppl 1:i14-i17. doi:10.1136/tobaccocontrol-2012-050860.
- 34. Donny EC, Hatsukami DK, Benowitz NL, Sved AF, Tidey JW, Cassidy RN. Reduced nicotine product standards for combustible tobacco: building an empirical basis for effective regulation. *Prev Med*. 2014;68:17-22. doi:10.1016/j.ypmed.2014.06.020.
- 35. Fagan P, King G, Lawrence D, et al. Eliminating tobacco-related health disparities: directions for future research. *Am J Public Health*. 2004;94(2):211-217.
- 36. Becker KM, Rose JE, Albino AP. A randomized trial of nicotine replacement therapy in combination with reduced-nicotine cigarettes for smoking cessation. *Nicotine Tob Res.* 2008;10(7):1139-1148. doi:10.1080/14622200802123294.
- 37. Benowitz NL, Hall SM, Stewart S, Wilson M, Dempsey D, Jacob P. Nicotine and carcinogen exposure with smoking of progressively reduced nicotine content cigarette. *Cancer Epidemiol Biomarkers Prev.* 2007;16(11):2479-2485. doi:10.1158/1055-9965.EPI-07-0393.
- 38. Benowitz NL, Dains KM, Hall SM, et al. Smoking behavior and exposure to tobacco toxicants during 6 months of smoking progressively reduced nicotine content cigarettes. *Cancer Epidemiol Biomarkers Prev*. 2012;21(5):761-769. doi:10.1158/1055-9965.EPI-11-0644.



- 39. Donny EC, Jones M. Prolonged exposure to denicotinized cigarettes with or without transdermal nicotine. *Drug Alcohol Depend*. 2009;104(1-2):23-33. doi:10.1016/j.drugalcdep.2009.01.021.
- 40. Donny EC, Houtsmuller E, Stitzer ML. Smoking in the absence of nicotine: behavioral, subjective and physiological effects over 11 days. *Addiction*. 2007;102(2):324-334. doi:10.1111/j.1360-0443.2006.01670.x.
- 41. Donny EC, Denlinger RL, Tidey JW, et al. Randomized trial of reduced-nicotine standards for cigarettes. *N Engl J Med*. 2015;373(14):1340-1349. doi:10.1056/NEJMsa1502403.
- 42. Hatsukami DK, Kotlyar M, Hertsgaard LA, et al. Reduced nicotine content cigarettes: effects on toxicant exposure, dependence and cessation. *Addiction*. 2010;105(2):343-355. doi:10.1111/j.1360-0443.2009.02780.x.
- 43. Hatsukami DK, Perkins KA, Lesage MG, et al. Nicotine reduction revisited: science and future directions. *Tob Control*. 2010;19(5):e1-e10. doi:10.1136/tc.2009.035584.
- 44. Hatsukami DK, Luo X, Dick L, et al. Reduced nicotine content cigarettes and use of alternative nicotine products: exploratory trial. *Addiction*. 2017;112(1):156-167. doi:10.1111/add.13603.
- 45. Walker N, Howe C, Bullen C, et al. The combined effect of very low nicotine content cigarettes, used as an adjunct to usual Quitline care (nicotine replacement therapy and behavioural support), on smoking cessation: a randomized controlled trial. *Addiction*. 2012;107(10):1857-1867. doi:10.1111/j.1360-0443.2012.03906.x.
- 46. Zeller M, Hatsukami D, Strategic dialogue on tobacco harm reduction group. The strategic dialogue on tobacco harm reduction: a vision and blueprint for action in the US. *Tob Control*. 2009;18(4):324-332. doi:10.1136/tc.2008.027318.
- 47. Dani JA, Harris RA. Nicotine addiction and comorbidity with alcohol abuse and mental illness. *Nat Neurosci*. 2005;8(11):1465-1470. doi:10.1038/nn1580.
- 48. Benowitz, N. Compensatory smoking of low-yield cigarettes. In: Shopland, Burns, Benowitz, Amacher, editors. NCI smoking and tobacco control monograph 13: Risks associated with smoking cigarettes with low machine-measured yields of tar and nicotine. Bethesda, MD: US Dept of Health and Human Services, Public Health Service, National Institutes of Health, National Cancer Institute; 2001. p 39-64.
- 49. Kozlowski LT, O'Connor RJ, Sweeney CT. Cigarette design. In: Shopland, Burns, Benowitz, Amacher, editors. NCI smoking and tobacco control monograph 13: Risks associated with smoking cigarettes with low machine-measured yields of tar and nicotine. Bethesda, MD: US Dept of Health and Human Services, Public Health Service, National Institutes of Health, National Cancer Institute; 2001. p 13-37.



- 50. Higgins ST, Heil SH, Sigmon SC, et al. Addiction potential of reduced nicotine content cigarettes in populations with psychiatric disorders and other vulnerabilities to tobacco addiction. *JAMA Psychiatry*. In press.
- Donny EC, Walker N, Hatsukami D, Bullen C. Reducing the nicotine content of combusted tobacco products sold in New Zealand. *Tob Control*. 2017;26(e1):e37e42. doi:10.1136/tobaccocontrol-2016-053186.
- 52. Benowitz NL, Donny EC, Hatsukami DK. Reduced nicotine content cigarettes, ecigarettes and the cigarette end game. *Addiction*. 2017;112(1):6-7. doi:10.1111/add.13534.
- 53. Quisenberry AJ, Koffarnus MN, Hatz LE, Epstein LH, Bickel WK. The Experimental Tobacco Marketplace I: Substitutability as a function of the price of conventional cigarettes. *Nicotine Tob Res.* 2016;18(7):1642-1648. doi:10.1093/ntr/ntv230.
- 54. Dawkins L, Kimber C, Puwanesarasa Y, Soar K. First- versus second-generation electronic cigarettes: predictors of choice and effects on urge to smoke and withdrawal symptoms. *Addiction*. 2015;110(4):669-677. doi:10.1111/add.12807.
- 55. Farsalinos KE, Spyrou A, Tsimopoulou K, Stefopoulos C, Romagna G, Voudris V. Nicotine absorption from electronic cigarette use: comparison between first and new-generation devices. *Sci Rep.* 2014;4:4133. doi:10.1038/srep04133.
- 56. Goniewicz ML, Kuma T, Gawron M, Knysak J, Kosmider L. Nicotine levels in electronic cigarettes. *Nicotine Tob Res.* 2013;15(1):158-166. doi:10.1093/ntr/nts103.
- 57. Talih S, Balhas Z, Eissenberg T, et al. Effects of user puff topography, device voltage, and liquid nicotine concentration on electronic cigarette nicotine yield: measurements and model predictions. *Nicotine Tob Res.* 2015;17(2):150-157. doi:10.1093/ntr/ntu174.
- 58. Trtchounian A, Williams M, Talbot P. Conventional and electronic cigarettes (ecigarettes) have different smoking characteristics. *Nicotine Tob Res.* 2010;12(9):905-912. doi:10.1093/ntr/ntq114.
- 59. Hecht SS, Carmella SG, Kotandeniya D, et al. Evaluation of toxicant and carcinogen metabolites in the urine of e-cigarette users versus cigarette smokers. *Nicotine Tob Res.* 2015;17(6):704-709. doi:10.1093/ntr/ntu218.
- 60. Goniewicz ML, Gawron M, Smith DM, Peng M, Jacob P, Benowitz NL. Exposure to nicotine and selected toxicants in cigarette smokers who switched to electronic cigarettes: A longitudinal within-subjects observational study. *Nicotine Tob Res*. 2017;19(2):160-167. doi:10.1093/ntr/ntw160.
- 61. Hefner K, Rosenheck R, Merrel J, Coffman M, Valentine G, Sofuoglu M. E-cigarette



- use in veterans seeking mental health and/or substance use services. *J Dual Diagn*. 2016;12(2):109-117. doi:10.1080/15504263.2016.1172895.
- 62. Hefner K, Valentine G, Sofuoglu M. Electronic cigarettes and mental illness: Reviewing the evidence for help and harm among those with psychiatric and substance use disorders. *Am J Addict*. 2017;26(4):306-315. doi:10.1111/ajad.12504.
- 63. Peters EN, Harrell PT, Hendricks PS, O'Grady KE, Pickworth WB, Vocci FJ. Electronic cigarettes in adults in outpatient substance use treatment: Awareness, perceptions, use, and reasons for use. *Am J Addict*. 2015;24(3):233-239. doi:10.1111/ajad.12206.
- 64. Prochaska JJ, Grana RA. E-cigarette use among smokers with serious mental illness. *PLoS ONE*. 2014;9(11):e113013. doi:10.1371/journal.pone.0113013.
- 65. Stein MD, Caviness CM, Grimone K, Audet D, Borges A, Anderson BJ. E-cigarette knowledge, attitudes, and use in opioid dependent smokers. *J Subst Abuse Treat*. 2015;52:73-77. doi:10.1016/j.jsat.2014.11.002.
- 66. Bullen C, Howe C, Laugesen M, et al. Electronic cigarettes for smoking cessation: a randomised controlled trial. *Lancet*. 2013;382(9905):1629-1637. doi:10.1016/S0140-6736(13)61842-5.
- 67. Caponnetto P, Auditore R, Russo C, Cappello GC, Polosa R. Impact of an electronic cigarette on smoking reduction and cessation in schizophrenic smokers: a prospective 12-month pilot study. *Int J Environ Res Public Health*. 2013;10(2):446-461. doi:10.3390/ijerph10020446.
- 68. Tseng T-Y, Ostroff JS, Campo A, et al. A randomized trial comparing the effect of nicotine versus placebo electronic cigarettes on smoking reduction among young adult smokers. *Nicotine Tob Res.* 2016;18(10):1937-1943. doi:10.1093/ntr/ntw017.
- 69. Adriaens K, Van Gucht D, Declerck P, Baeyens F. Effectiveness of the electronic cigarette: An eight-week Flemish study with six-month follow-up on smoking reduction, craving and experienced benefits and complaints. *Int J Environ Res Public Health*. 2014;11(11):11220-11248. doi:10.3390/ijerph111111220.
- 70. Stein MD, Caviness C, Grimone K, Audet D, Anderson BJ, Bailey GL. An open trial of electronic cigarettes for smoking cessation among methadone-maintained smokers. *Nicotine Tob Res.* 2016;18(5):1157-1162. doi:10.1093/ntr/ntv267.
- 71. Glasser AM, Collins L, Pearson JL, et al. Overview of electronic nicotine delivery systems: A systematic review. *Am J Prev Med*. 2017;52(2):e33-e66. doi:10.1016/j.amepre.2016.10.036.



- 72. Lechner WV, Meier E, Wiener JL, et al. The comparative efficacy of first- versus second-generation electronic cigarettes in reducing symptoms of nicotine withdrawal. *Addiction*. 2015;110(5):862-867. doi:10.1111/add.12870.
- 73. Vansickel AR, Eissenberg T. Electronic cigarettes: effective nicotine delivery after acute administration. *Nicotine Tob Res.* 2013;15(1):267-270. doi:10.1093/ntr/ntr316.
- 74. Bonhomme MG, Holder-Hayes E, Ambrose BK, et al. Flavoured non-cigarette tobacco product use among US adults: 2013-2014. *Tob Control*. 2016;25(Suppl 2):ii4-ii13. doi:10.1136/tobaccocontrol-2016-053373.
- 75. Audrain-McGovern J, Strasser AA, Wileyto EP. The impact of flavoring on the rewarding and reinforcing value of e-cigarettes with nicotine among young adult smokers. *Drug Alcohol Depend*. 2016;166:263-267. doi:10.1016/j.drugalcdep.2016.06.030.
- 76. Goldenson NI, Kirkpatrick MG, Barrington-Trimis JL, et al. Effects of sweet flavorings and nicotine on the appeal and sensory properties of e-cigarettes among young adult vapers: Application of a novel methodology. *Drug Alcohol Depend*. 2016;168:176-180. doi:10.1016/j.drugalcdep.2016.09.014.
- 77. Berg CJ. Preferred flavors and reasons for e-cigarette use and discontinued use among never, current, and former smokers. *Int J Public Health*. 2016;61(2):225-236. doi:10.1007/s00038-015-0764-x.
- 78. Kistler CE, Crutchfield TM, Sutfin EL, et al. Consumers' preferences for electronic nicotine delivery system product features: A structured content analysis. *Int J Environ Res Public Health*. 2017;14(6). doi:10.3390/ijerph14060613.
- 79. Czoli CD, Goniewicz M, Islam T, Kotnowski K, Hammond D. Consumer preferences for electronic cigarettes: results from a discrete choice experiment. *Tob Control*. 2016;25(e1):e30-e36. doi:10.1136/tobaccocontrol-2015-052422.
- 80. Pesko MF, Kenkel DS, Wang H, Hughes JM. The effect of potential electronic nicotine delivery system regulations on nicotine product selection. *Addiction*. 2016;111(4):734-744. doi:10.1111/add.13257.
- 81. Etter JF. Electronic cigarettes: a survey of users. *BMC Public Health*. 2010;10:231. doi:10.1186/1471-2458-10-231.
- 82. Farsalinos KE, Romagna G, Tsiapras D, Kyrzopoulos S, Spyrou A, Voudris V. Impact of flavour variability on electronic cigarette use experience: an internet survey. *Int J Environ Res Public Health*. 2013;10(12):7272-7282. doi:10.3390/ijerph10127272.



- 83. Litt MD, Duffy V, Oncken C. Cigarette smoking and electronic cigarette vaping patterns as a function of e-cigarette flavourings. *Tob Control*. 2016;25(Suppl 2):ii67-ii72. doi:10.1136/tobaccocontrol-2016-053223.
- 84. Yingst JM, Veldheer S, Hrabovsky S, Nichols TT, Wilson SJ, Foulds J. Factors associated with electronic cigarette users' device preferences and transition from first generation to advanced generation devices. *Nicotine Tob Res.* 2015;17(10):1242-1246. doi:10.1093/ntr/ntv052.
- 85. Bogucka-Bonikowska A, Baran-Furga H, Chmielewska K, et al. Taste function in methadone-maintained opioid-dependent men. *Drug Alcohol Depend*. 2002;68(1):113-117.
- 86. Fenn JM, Laurent JS, Sigmon SC. Increases in body mass index following initiation of methadone treatment. *J Subst Abuse Treat*. 2015;51:59-63. doi:10.1016/j.jsat.2014.10.007.
- 87. Mysels DJ, Sullivan MA. The relationship between opioid and sugar intake: review of evidence and clinical applications. *J Opioid Manag*. 2010;6(6):445-452.
- 88. Nolan LJ, Scagnelli LM. Preference for sweet foods and higher body mass index in patients being treated in long-term methadone maintenance. *Subst Use Misuse*. 2007;42(10):1555-1566. doi:10.1080/10826080701517727.
- 89. Olszewski PK, Levine AS. Central opioids and consumption of sweet tastants: when reward outweighs homeostasis. *Physiol Behav*. 2007;91(5):506-512. doi:10.1016/j.physbeh.2007.01.011.
- 90. Zador D, Lyons Wall PM, Webster I. High sugar intake in a group of women on methadone maintenance in south western Sydney, Australia. *Addiction*. 1996;91(7):1053-1061.
- 91. Chait LD, Griffiths RR. Effects of methadone on human cigarette smoking and subjective ratings. *J Pharmacol Exp Ther*. 1984;229(3):636-640.
- 92. Higgins ST, Budney AJ, Hughes JR, Bickel WK, Lynn M, Mortensen A. Influence of cocaine use on cigarette smoking. *JAMA*. 1994;272(22):1724.
- 93. Mello NK, Mendelson JH, Sellers ML, Kuehnle JC. Effects of heroin self-administration on cigarette smoking. *Psychopharmacology (Berl)*. 1980;67(1):45-52.
- 94. Mello NK, Lukas SE, Mendelson JH. Buprenorphine effects on cigarette smoking. *Psychopharmacology (Berl)*. 1985;86(4):417-425.
- 95. Roll JM, Higgins ST, Tidey J. Cocaine use can increase cigarette smoking: evidence from laboratory and naturalistic settings. *Exp Clin Psychopharmacol*.



- 1997;5(3):263-268.
- 96. Schmitz JM, Grabowski J, Rhoades H. The effects of high and low doses of methadone on cigarette smoking. *Drug Alcohol Depend*. 1994;34(3):237-242.
- 97. Dunn KE, Sigmon SC, Thomas CS, Heil SH, Higgins ST. Voucher-based contingent reinforcement of smoking abstinence among methadone-maintained patients: a pilot study. *J Appl Behav Anal*. 2008;41(4):527-538.
- 98. Dunn KE, Sigmon SC, Reimann EF, Badger GJ, Heil SH, Higgins ST. A contingency-management intervention to promote initial smoking cessation among opioid-maintained patients. *Exp Clin Psychopharmacol*. 2010;18(1):37-50. doi:10.1037/a0018649.
- 99. Sigmon SC, Miller ME, Meyer AC, et al. Financial incentives to promote extended smoking abstinence in opioid-maintained patients: a randomized trial. *Addiction*. 2016;111(5):903-912. doi:10.1111/add.13264.
- 100. Higgins ST, Heil SH, Sigmon SC, et al. Response to varying the nicotine content of cigarettes in vulnerable populations: an initial experimental examination of acute effects. *Psychopharmacology (Berl)*. 2017;234(1):89-98. doi:10.1007/s00213-016-4438-z.
- 101. Beck AT, Steer RA, Brown GK. Manual for Beck Depression Inventory II 1996; San Antonio, TX: Psychological Corporation.
- 102. Norman SB, Cissell SH, Means-Christensen AJ, Stein MB. Development and validation of an Overall Anxiety Severity And Impairment Scale (OASIS). Depress Anxiety. 2006;23(4):245-249.
- 103. Sheehan DV, Lecrubier Y, Sheehan KH, et al. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33.
- 104. Sheehan DV, Lecrubier Y, Sheehan K, Harnett, Janavs J, Weiller E, et al. (1997). The validity of the Mini International Neuropsychiatric Interview (MINI) according to the SCID-P and its reliability. *Eur Psychiat 12*, 232–241.
- 105. Babor TF, de la Fuente JR, Saunders J, Grant M. AUDIT: The Alcohol Use Disorders Identification Test.Guidelines for use in primary health care. Geneva: World Health Organization, 1992.
- 106. Skinner HA. The Drug Abuse Screening Test. Addict Behav. 1982; 7(4):363-371.
- 107. Heatherton TF, Kozlowski LT, Frecker RC, Fagerström KO. The Fagerström Test for Nicotine Dependence: a revision of the Fagerström Tolerance Questionnaire. Br J Addict. 1991;86(9):1119-1127.



- 108. Piper ME, McCarthy DE, Bolt DM, Smith SS, Lerman C, Benowitz N, et al. Assessing dimensions of nicotine dependence: An evaluation of the Nicotine Dependence Syndrome Scale (NDSS) and the Wisconsin Inventory of Smoking Dependence Motives (WISDM) Nicotine & Tobacco Research. 2008;10:1009–1020.
- 109. Foulds J, Veldheer S, Yingst J, Wilson SJ, Nichols TT, Eissenberg T. Development of a questionnaire for assessing dependence on electronic cigarettes among a large sample of ex-smoking E-cigarette users. Nicotine Tob Res. 2015; 17(2): 186-92.
- 110. DiClemente CC, Prochaska JO, Fairhurst SK, Velicer WF, Velasquez MM, Rossi JS. The process of smoking cessation: an analysis of precontemplation, contemplation, and preparation stages of change. J Consult Clin Psychol. 1991;59(2):295-304.
- 111. McLellan ST, Luborsky L, Cacciola J, Griffith JE, Evans F, Barr HL, O'Brien CP. New data from the Addiction Severity Index: Reliability and validity in three centers. Journal of Nervous and Mental Disease. 1985;173:412-423.
- 112. Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983;24(4):385-396.
- 113. Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988;54(6):1063-1070.
- 114. Hughes JR, Hatsukami D. Signs and symptoms of tobacco withdrawal. Arch Gen Psychiatry. 1986;43(3):289-294.
- 115. Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001;3(1):7-16.
- 116. Dowd AN, Motschman CA, Tiffany ST. Development and Validation of the Questionnaire of Vaping Craving. Nicotine Tob Res. 2019;12(1):63-70.
- 117. Cappelleri JC, Bushmakin AG, Baker CL, Merikle E, Olufade AO, Gilbert DG. Confirmatory factor analyses and reliability of the modified cigarette evaluation questionnaire. Addict Behav. 2007;32(5):912-923.
- 118. Jacobs EA, Bickel WK. Modeling drug consumption in the clinic using simulation procedures: demand for heroin and cigarettes in opioid-dependent outpatients. Exp Clin Psychopharmacol. 1999;7(4):412-426.
- 119. Cassidy RN, Tidey JW, Colby SM, Long V, Higgins ST. Initial development of an ecigarette purchase task: a mixed methods study. Tob Regul Sci. 2017; 3(2): 139-150.
- 120. Grace RC, Kivel BM, Laugesen M. Estimating cross-price elasticity of e-cigarettes using a simulated demand procedure. Nicotine Tob Res. 2015 May;17(5):592-598.



121. Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith–Hamilton Pleasure Scale. British Journal of Psychiatry. 1995;167:99–103.